CLINICAL TRIAL: NCT05374525
Title: A Phase 4, Randomized, Open-label, Two-arm Study Evaluating Implementation Strategies for the Delivery of Cabotegravir in Low and High-volume Pre-exposure Prophylaxis (PrEP) Sites in the U.S. for HIV Uninfected MSM and Transgender Men ≥ 18
Brief Title: A Study Evaluating Implementation Strategies for the Delivery of Cabotegravir in Low and High-Volume PrEP Site in the United States
Acronym: PILLAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 217710
Expanded Access: NCT03462810 (Available)
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections
Keywords: Cabotegravir; Long-acting injectables; Implementation science; HIV; Pre-exposure prophylaxis
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dynamic Implementation (DI) - PSP (Experimental): Men who have sex with men (MSM) and transgender men (TGM) who were HIV negative as PSPs received APRETUDE injection (Direct to Injection - DTI) and had the choice to receive an optional cabotegravir tablets as oral lead in (OLI). PSPs had access to enhanced toolkits and digital health implementation supports.
  Interventions: Drug: APRETUDE; Drug: Cabotegravir OLI
- Routine Implementation (RI) - PSP (Experimental): MSM and transgender men who were HIV negative as PSPs received APRETUDE injection (DTI) and had the choice to use an optional cabotegravir tablets as OLI. PSPs had access to standard toolkits for APRETUDE to use as needed.
  Interventions: Drug: APRETUDE; Drug: Cabotegravir OLI

INTERVENTIONS:
Drug: APRETUDE — Available as intramuscular injection.
Drug: Cabotegravir OLI — Available as marketed orally administered tablets.

SUMMARY:
This is a two-arm study evaluating the impact of two implementation strategy conditions, dynamic implementation and routine implementation on the feasibility of delivering of Cabotegravir PrEP in low and high-volume PrEP sites in the United States for men who have sex with men (MSM) and Transgender men ≥ 18 years of age. There are two types of participants in the study. Patient Study Participants (PSPs) will refer to individuals who are enrolled in the study and who will receive commercially available Cabotegravir PrEP via prescription from the PrEP provider at the corresponding site. Staff Study Participants (SSPs) will refer to site staff who are involved in administrative and clinical aspects of offering and administering PrEP to PSPs and will participate in the staff study assessments. PSPs who choose to opt for 1-month oral lead-in (OLI) will receive cabotegravir tablets for PrEP at Month 1 followed by APPRETUDE intramuscular (IM) injections on Month 2, 3 and every two months thereafter up to Month 13. PSPs who opt for Direct to injections (DTI) will receive APPRETUDE IM injections on Month 1, 2 and every two months thereafter up to Month 12. Month 6/7 refers to Month 6 (DTI)/ Month 7 (OLI). Month 12/13 refers to Month 12 (DTI)/ Month 13 (OLI).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age inclusive, at the time of signing the informed consent.
* No prior history of receiving CAB PrEP
* HIV negative test result at screening
* Capable of giving signed informed consent form

Exclusion Criteria:

* HIV indeterminate or positive test result during screening and prior to initiation of CAB PrEP
* A participant of concurrent interventional clinical or implementation science study at any time during the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men who have sex with Men or Transgender Men
Enrollment: 287 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (17):
- United States (17):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Bridgeport, Kansas
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Harlingen, Texas
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 Clinics were randomized to Dynamic Implementation and Routine Implementation arms. In these clinics, a total of 201 patient study participants (PSPs) were enrolled in the study and all of them received study treatment and 86 Staff Study Participants (SSPs) were enrolled that included healthcare providers, nurses, staff performing injections, clinic administrators, pharmacists and laboratory staff.
Pre-assignment Details: SSPs provided input through surveys and semi-structured interviews. Baseline characteristics and adverse events for SSP were not collected as it was not required per study design.
Units Other Than Participants: Clinics
Groups:
- Dynamic Implementation (DI): The DI arm evaluated the feasibility of APRETUDE delivery with implementation supports. Clinics randomized to DI received enhanced toolkits, a digital health end to end implementation strategy; and implementation facilitation.
- Routine Implementation (RI): The RI arm evaluated the feasibility of APRETUDE delivery without implementation supports. Sites randomized to RI had access to the standard toolkits for SSPs and PSPs that were available for APRETUDE to use as needed.
Period: Overall Study
Arm/Group | Dynamic Implementation (DI) | Routine Implementation (RI)
Started | 173; 11 Clinics | 114; 6 Clinics
PSP | 117; 11 Clinics | 84; 6 Clinics
SSP | 56; 11 Clinics | 30; 6 Clinics
Completed | 137; 11 Clinics | 95; 6 Clinics
Not Completed | 36; 0 Clinics | 19; 0 Clinics
Not completed — Adverse Event | 5 | 6
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 2 | 2
Not completed — Withdrawal by Subject | 26 | 8

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for SSPs were not collected as it was not required as per study design.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP | Total
Number analyzed (Participants) | 117 | 84 | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.6 (11.16) | 37.8 (10.76) | 37.7 (10.97)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Self-identified gender data at the time of enrollment is reported.
  Participants
    Cisgender Man | 107 | 82 | 189
    Transgender Man | 10 | 2 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 2 | 8
  Black of African American | 19 | 29 | 48
  Multiple Races | 2 | 4 | 6
  Other, not specified | 2 | 0 | 2
  Unknown | 15 | 2 | 17
  White | 72 | 47 | 119

OUTCOME MEASURES:

1. Primary Outcome: Mean Feasibility of Intervention Measure (FIM) Score Assessed for SSPs
Description: The FIM-Intervention (INT) was a four-item measure for APRETUDE intervention (1. APRETUDE seems implementable in our clinic/practice 2. APRETUDE seems possible in our clinic/practice 3. APRETUDE seems doable in our clinic/practice 4. APRETUDE seems easy to use in our clinic/practice) and was measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least feasibility and 5 the most feasibility.
  Timeframe for evaluation of this outcome measure is Month (M)12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI)
Time Frame: At Month 12
Population: Analysis was performed on the SSPs who completed at least one survey at any time point. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- DI - SSP: Staff at sites offering APRETUDE injection for pre- exposure prophylaxis (PrEP). SSPs had access to enhanced toolkits, a digital health implementation strategy and implementation facilitation for APRETUDE.
- RI - SSP: Staff at sites offering APRETUDE injection for PrEP. SSPs had access to standard toolkits for APRETUDE to use as needed.
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 52 | 29
Scores on a scale | 4.37 (0.68) | 4.27 (0.68)

2. Secondary Outcome: Change From Baseline in FIM Score Assessed for SSPs
Description: This outcome assesses the change in FIM-INT for SSPs over time. The FIM-INT was a four-item measure for APRETUDE intervention (1. APRETUDE seems implementable in our clinic/practice 2. APRETUDE seems possible in our clinic/practice 3. APRETUDE seems doable in our clinic/practice 4. APRETUDE seems easy to use in our clinic/practice) and was measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least feasibility and 5 the most feasibility.
  Timeframe for evaluation of this outcome measure is M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI) compared to Baseline (BL).
Time Frame: At Month 4 and Month 12 compared to baseline (Month 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 48 | 29
Scores on a scale
  Month 4 compared to baseline (BL) | -0.29 (0.92) | 0.08 (0.59)
  Month 12 compared to BL: number analyzed (Participants) | 40 | 26
  Month 12 compared to BL | -0.01 (0.69) | -0.11 (0.86)

3. Secondary Outcome: Number of SSPs Assessed for Perceptions of Facilitators to RI, DI and Overall Implementation of PrEP Into Routine Care Through Month 12
Description: Perception of facilitators to RI, DI and overall implementation of PrEP measured from themes emerging from Proctor and Consolidated Framework for Implementation Research (CFIR) guided semi-structured qualitative interviews. In this outcome measure, SSPs were asked about the facilitators of the overall implementation of APRETUDE into clinic infrastructure, evaluating feasibility of DI and RI study arms.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on the SSPs who were interviewed and had data available for the specified analysis at the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 14 | 10
Participants
  Clinic being flexible with scheduling (injection/ lab visits) | 5 | 1
  Scheduling appointments in advance | 6 | 0
  Training and consistent information provided to staff | 5 | 0
  Increased communication for vulnerable populations | 3 | 1
  Previous experience with CABENUVA/ APRETUDE | 2 | 2

4. Secondary Outcome: Number of SSPs Assessed for Perceptions of Barriers to RI, DI and Overall Implementation of PrEP Into Routine Care Through Month 12
Description: Perception of barriers to RI, DI and overall implementation of PrEP measured from themes emerging from Proctor and CFIR guided semi-structured qualitative interview. In this outcome measure, SSPs were asked about the barriers/challenges of the overall implementation of APRETUDE into clinic infrastructure, evaluating feasibility of DI and RI study arms.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 14 | 10
Participants
  Staff burden to integrate the new process | 7 | 3
  Complex team coordination | 4 | 2
  Insurance challenges related to infrastructure | 4 | 2
  Infrastructure Logistic challenges | 3 | 2
  Follow-up with pharmacies needed to obtain APRETUDE | 2 | 2

5. Secondary Outcome: Mean FIM Score Assessed for PSPs
Description: The FIM-INT was a four-item measure for APRETUDE intervention (1. Receiving APRETUDE injection every 2 months seems workable in my life 2. Receiving APRETUDE injection every 2 months seems possible in my life 3. Receiving APRETUDE injection every 2 months seems doable in my life 4. Receiving APRETUDE injection every 2 months seems easy in my life) and was measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least feasibility and 5 the most feasibility.
  Timeframe for evaluation of this outcome measure is BL, M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Baseline (Month 1), Month 6 and Month 12
Population: Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who successfully completed a portion of the survey. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 105 | 77
Scores on a scale
  Baseline | 4.33 (0.77) | 4.51 (0.70)
  Month 6: number analyzed (Participants) | 94 | 65
  Month 6 | 4.35 (0.75) | 4.46 (0.73)
  Month 12: number analyzed (Participants) | 77 | 63
  Month 12 | 4.36 (0.79) | 4.46 (0.72)

6. Secondary Outcome: Mean Acceptability of Intervention Measure (AIM) Score Assessed for PSPs
Description: The AIM-INT was employed to evaluate the perceived intervention acceptability among PSPs. The measure consists of four items (1. APRETUDE meets my approval for preventing HIV 2. APRETUDE for the prevention of HIV is appealing to me 3. I like APRETUDE for the prevention of HIV 4. I welcome APRETUDE for the prevention of HIV), each with a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least acceptability and 5 the most acceptability.
  Timeframe for evaluation of this outcome measure is BL, M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Baseline (Month 1), Month 6 and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 105 | 77
Scores on a scale
  Baseline | 4.46 (0.69) | 4.41 (0.68)
  Month 6: number analyzed (Participants) | 94 | 65
  Month 6 | 4.57 (0.64) | 4.57 (0.55)
  Month 12: number analyzed (Participants) | 77 | 63
  Month 12 | 4.61 (0.63) | 4.60 (0.67)

7. Secondary Outcome: Number of PSPs With Responses to Implementation Science Questionnaire (ISQ) Regarding Their Feelings About Taking APRETUDE
Description: The implementation science questionnaire (ISQ) used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs indicated their feelings about taking APRETUDE.
  Timeframe for evaluation of this outcome measure is BL, M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Baseline (Month 1), Month 6 and Month 12
Population: Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who completed at least one ISQ survey at any timepoint. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  At Baseline - Overall, how are you feeling about taking APRETUDE?: Very Positive | 79 | 64
  At Baseline - Overall, how are you feeling about taking APRETUDE?: Somewhat Positive | 19 | 10
  At Baseline - Overall, how are you feeling about taking APRETUDE?: Neither positive nor negative | 7 | 1
  At Baseline - Overall, how are you feeling about taking APRETUDE?: Somewhat negative | 0 | 0
  At Baseline - Overall, how are you feeling about taking APRETUDE?: Very negative | 0 | 0
  At Baseline - Overall, how are you feeling about taking APRETUDE?: Missing | 12 | 9
  At Month 6 - Overall, how are you feeling about taking APRETUDE?: Very Positive | 72 | 52
  At Month 6 - Overall, how are you feeling about taking APRETUDE?: Somewhat Positive | 16 | 9
  At Month 6 - Overall, how are you feeling about taking APRETUDE?: Neither positive nor negative | 2 | 1
  At Month 6 - Overall, how are you feeling about taking APRETUDE?: Somewhat negative | 2 | 1
  At Month 6 - Overall, how are you feeling about taking APRETUDE?: Very negative | 0 | 0
  At Month 6 - Overall, how are you feeling about taking APRETUDE?: Missing | 25 | 21
  At Month 12 - Overall, how are you feeling about taking APRETUDE?: Very Positive | 66 | 55
  At Month 12 - Overall, how are you feeling about taking APRETUDE?: Somewhat Positive | 10 | 7
  At Month 12 - Overall, how are you feeling about taking APRETUDE?: Neither positive nor negative | 0 | 1
  At Month 12 - Overall, how are you feeling about taking APRETUDE?: Somewhat negative | 1 | 0
  At Month 12 - Overall, how are you feeling about taking APRETUDE?: Very negative | 0 | 0
  At Month 12 - Overall, how are you feeling about taking APRETUDE?: Missing | 40 | 21

8. Secondary Outcome: Number of PSPs With Responses to ISQs Regarding Acceptability of Coming to Clinic for APRETUDE Injection
Description: The ISQ used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs indicated how acceptable it was for them to go to the clinic for APRETUDE injections.
  Timeframe for evaluation of this outcome measure is BL, M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Baseline (Month 1), Month 6 and Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  At Baseline - How acceptable is coming to the clinic every 2 months for an injection?: Very acceptable | 60 | 55
  At Baseline - How acceptable is coming to the clinic every 2 months for an injection?: Acceptable | 31 | 19
  At Baseline - How acceptable is coming to the clinic every 2 months for an injection?: Somewhat acceptable | 10 | 2
  At Baseline - How acceptable is coming to the clinic every 2 months for an injection?: A little acceptable | 4 | 0
  At Baseline - How acceptable is coming to the clinic every 2 months for an injection?: Not at all acceptable | 0 | 0
  At Baseline - How acceptable is coming to the clinic every 2 months for an injection?: Missing | 12 | 8
  At Month 6 - How acceptable is coming to the clinic every 2 months for an injection?: number analyzed (Participants) | 92 | 63
  At Month 6 - How acceptable is coming to the clinic every 2 months for an injection?: Very acceptable | 49 | 40
  At Month 6 - How acceptable is coming to the clinic every 2 months for an injection?: Acceptable | 31 | 16
  At Month 6 - How acceptable is coming to the clinic every 2 months for an injection?: Somewhat acceptable | 8 | 6
  At Month 6 - How acceptable is coming to the clinic every 2 months for an injection?: A little acceptable | 3 | 0
  At Month 6 - How acceptable is coming to the clinic every 2 months for an injection?: Not at all acceptable | 1 | 1
  At Month 6 - How acceptable is coming to the clinic every 2 months for an injection?: Missing | 0 | 0
  At Month 12 - How acceptable is coming to the clinic every 2 months for an injection?: number analyzed (Participants) | 76 | 63
  At Month 12 - How acceptable is coming to the clinic every 2 months for an injection?: Very acceptable | 41 | 39
  At Month 12 - How acceptable is coming to the clinic every 2 months for an injection?: Acceptable | 21 | 18
  At Month 12 - How acceptable is coming to the clinic every 2 months for an injection?: Somewhat acceptable | 11 | 5
  At Month 12 - How acceptable is coming to the clinic every 2 months for an injection?: A little acceptable | 3 | 1
  At Month 12 - How acceptable is coming to the clinic every 2 months for an injection?: Not at all acceptable | 0 | 0
  At Month 12 - How acceptable is coming to the clinic every 2 months for an injection?: Missing | 0 | 0

9. Secondary Outcome: Number of PSPs With Responses to the ISQs Regarding Recommending APRETUDE
Description: The ISQ used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs indicated if they would recommend APRETUDE to others.
  Timeframe for evaluation of this outcome measure is M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Month 6 and Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  At Month 6 - I would recommend APRETUDE to other people who could benefit from it: Completely agree | 72 | 49
  At Month 6 - I would recommend APRETUDE to other people who could benefit from it: Agree | 18 | 12
  At Month 6 - I would recommend APRETUDE to other people who could benefit from it: Neither agree nor disagree | 2 | 0
  At Month 6 - I would recommend APRETUDE to other people who could benefit from it: Disagree | 0 | 1
  At Month 6 - I would recommend APRETUDE to other people who could benefit from it: Completely disagree | 0 | 1
  At Month 6 - I would recommend APRETUDE to other people who could benefit from it: Missing | 25 | 21
  At Month 12 - I would recommend APRETUDE to other people who could benefit from it: Completely agree | 64 | 52
  At Month 12 - I would recommend APRETUDE to other people who could benefit from it: Agree | 12 | 9
  At Month 12 - I would recommend APRETUDE to other people who could benefit from it: Neither agree nor disagree | 1 | 2
  At Month 12 - I would recommend APRETUDE to other people who could benefit from it: Disagree | 0 | 0
  At Month 12 - I would recommend APRETUDE to other people who could benefit from it: Completely disagree | 0 | 0
  At Month 12 - I would recommend APRETUDE to other people who could benefit from it: Missing | 40 | 21

10. Secondary Outcome: Number of PSPs With Responses to the ISQs Regarding Appointment Scheduling
Description: The ISQ used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs were asked about their opinion on the ease or difficulty of scheduling appointments at the clinic.
  Timeframe for evaluation of this outcome measure is M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Month 6 and Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  Month 6- How easy or difficult is it to schedule appointments for your injections?: Very easy | 60 | 46
  Month 6- How easy or difficult is it to schedule appointments for your injections?: Somewhat easy | 20 | 13
  Month 6- How easy or difficult is it to schedule appointments for your injections?: Neither easy nor difficult | 5 | 3
  Month 6- How easy or difficult is it to schedule appointments for your injections?: Somewhat difficult | 6 | 1
  Month 6- How easy or difficult is it to schedule appointments for your injections?: Very difficult | 2 | 0
  Month 6- How easy or difficult is it to schedule appointments for your injections?: I have not scheduled any appointments at the clinic/practice | 0 | 0
  Month 6- How easy or difficult is it to schedule appointments for your injections?: Missing | 24 | 21
  Month 12- How easy or difficult is it to schedule appointments for your injections?: Very easy | 49 | 46
  Month 12- How easy or difficult is it to schedule appointments for your injections?: Somewhat easy | 15 | 10
  Month 12- How easy or difficult is it to schedule appointments for your injections?: Neither easy nor difficult | 6 | 4
  Month 12- How easy or difficult is it to schedule appointments for your injections?: Somewhat difficult | 5 | 2
  Month 12- How easy or difficult is it to schedule appointments for your injections?: Very difficult | 1 | 1
  Month 12- How easy or difficult is it to schedule appointments for your injections?: I have not scheduled any appointments at the clinic/practice | 1 | 0
  Month 12- How easy or difficult is it to schedule appointments for your injections?: Missing | 40 | 21

11. Secondary Outcome: Number of PSPs With Responses to the ISQs Regarding Appointment Rescheduling
Description: The ISQ used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs were asked about their opinion on ease or difficulty of rescheduling appointments at the clinic.
  Timeframe for evaluation of this outcome measure is M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Month 6 and Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 93 | 63
Participants
  Month 6 - How easy or difficult is it to reschedule appointments for your injections?: Very easy | 44 | 25
  Month 6 - How easy or difficult is it to reschedule appointments for your injections?: Somewhat easy | 14 | 17
  Month 6 - How easy or difficult is it to reschedule appointments for your injections?: Neither easy nor difficult | 1 | 4
  Month 6 - How easy or difficult is it to reschedule appointments for your injections?: Somewhat difficult | 6 | 2
  Month 6 - How easy or difficult is it to reschedule appointments for your injections?: Very difficult | 3 | 1
  Month 6 - How easy or difficult is it to reschedule appointments for your injections?: I have not needed to reschedule any appointments | 25 | 14
  Month 12- How easy or difficult is it to reschedule appointments for your injections?: number analyzed (Participants) | 76 | 63
  Month 12- How easy or difficult is it to reschedule appointments for your injections?: Very easy | 39 | 30
  Month 12- How easy or difficult is it to reschedule appointments for your injections?: Somewhat easy | 13 | 17
  Month 12- How easy or difficult is it to reschedule appointments for your injections?: Neither easy nor difficult | 4 | 4
  Month 12- How easy or difficult is it to reschedule appointments for your injections?: Somewhat difficult | 8 | 6
  Month 12- How easy or difficult is it to reschedule appointments for your injections?: Very difficult | 2 | 1
  Month 12- How easy or difficult is it to reschedule appointments for your injections?: I have not needed to reschedule any appointments | 10 | 5

12. Secondary Outcome: Change From Baseline in AIM Score Assessed for PSPs
Description: This outcome assesses the change in AIM-INT for PSPs over time. The measure consists of four items (1. APRETUDE meets my approval for preventing HIV 2. APRETUDE for the prevention of HIV is appealing to me 3. I like APRETUDE for the prevention of HIV 4. I welcome APRETUDE for the prevention of HIV), each with a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least acceptability and 5 the most acceptability.
  Timeframe for evaluation of this outcome measure is M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI) compared to Baseline.
Time Frame: At Month 6 and Month 12 compared to baseline (Month 1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 87 | 61
Scores on a scale
  Month 6 compared to BL | 0.17 (0.66) | 0.20 (0.72)
  Month 12 compared to BL: number analyzed (Participants) | 71 | 59
  Month 12 compared to BL | 0.27 (0.63) | 0.19 (0.87)

13. Secondary Outcome: Change From Baseline in FIM Score Assessed for PSPs
Description: This outcome assesses the change in FIM-INT for PSPs over time. The FIM-INT was a four-item measure for APRETUDE intervention (1. Receiving APRETUDE injection every 2 months seems workable in my life 2. Receiving APRETUDE injection every 2 months seems possible in my life 3. Receiving APRETUDE injection every 2 months seems doable in my life 4. Receiving APRETUDE injection every 2 months seems easy in my life) and was measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least feasibility and 5 the most feasibility.
  Timeframe for evaluation of this outcome measure is M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI) compared to baseline.
Time Frame: At Month 6 and Month 12 compared to baseline (Month 1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 87 | 61
Scores on a scale
  Month 6 compared to BL | 0.01 (0.80) | 0.00 (0.89)
  Month 12 compared to BL: number analyzed (Participants) | 71 | 59
  Month 12 compared to BL | 0.01 (0.71) | -0.01 (0.92)

14. Secondary Outcome: Percentage of PSPs With Change From Baseline in ISQ Responses
Description: The ISQ used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs indicated their feelings about taking APRETUDE and how acceptable it was for them to go to the clinic for APRETUDE injections. Timeframe for evaluation of this outcome measure is BL, M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI). The change from baseline is calculated as a difference of percentages resulted at each timepoint as following: M6 minus (-) BL, and M12-BL. Q2M = a schedule of injection administration at every 2 months.
Time Frame: At Month 6 and Month 12 compared to Baseline (Month 1)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Groups:
- DI- PSP: Men who have sex with men (MSM) and transgender men (TGM) who were HIV negative as PSPs received APRETUDE injection (Direct to Injection - DTI) and had the choice to receive an optional cabotegravir tablets as oral lead in (OLI). PSPs had access to enhanced toolkits and digital health implementation supports.
- RI- PSP: MSM and transgender men who were HIV negative as PSPs received APRETUDE injection (DTI) and had the choice to use an optional cabotegravir tablets as OLI. PSPs had access to standard toolkits for APRETUDE to use as needed.
Arm/Group | DI- PSP | RI- PSP
Number analyzed (Participants) | 92 | 63
Percentage of participants
  Change BL to M6 - How the participant felt about taking APRETUDE - Very positive | 3.0 | -2.8
  Change BL to M6 - How the participant felt about taking APRETUDE - Somewhat positive | -0.7 | 1.0
  Change BL to M6-How the participant felt about taking APRETUDE- Neither positive nor negative | -4.5 | 0.3
  Change BL to M6 - How the participant felt about taking APRETUDE - Somewhat negative | 2.2 | 1.6
  Change BL to M6 - How the participant felt about taking APRETUDE - Very negative | 0.0 | 0.0
  Change BL to M12 - How the participant felt about taking APRETUDE-Very positive: number analyzed (Participants) | 77 | 63
  Change BL to M12 - How the participant felt about taking APRETUDE-Very positive | 10.5 | 2.0
  Change BL to M12 - How the participant felt about taking APRETUDE-Somewhat positive: number analyzed (Participants) | 77 | 63
  Change BL to M12 - How the participant felt about taking APRETUDE-Somewhat positive | -5.1 | -2.2
  Change BL to M12-How the participant felt about taking APRETUDE-Neither positive nor negative: number analyzed (Participants) | 77 | 63
  Change BL to M12-How the participant felt about taking APRETUDE-Neither positive nor negative | -6.7 | 0.3
  Change BL to M12 - How the participant felt about taking APRETUDE-Somewhat negative: number analyzed (Participants) | 77 | 63
  Change BL to M12 - How the participant felt about taking APRETUDE-Somewhat negative | 1.3 | 0.0
  Change BL to M12 - How the participant felt about taking APRETUDE-Very negative: number analyzed (Participants) | 77 | 63
  Change BL to M12 - How the participant felt about taking APRETUDE-Very negative | 0.0 | 0.0
  Change BL to M6 - Participant' acceptability for injection visits Q2M - Very acceptable | -3.9 | -8.9
  Change BL to M6 - Participant' acceptability for injection visits Q2M - Acceptable | 4.2 | 0.4
  Change BL to M6 - Participant' acceptability for injection visits Q2M - Somewhat acceptable | -0.8 | 6.9
  Change BL to M6 - Participant' acceptability for injection visits Q2M - A little acceptable | -0.5 | 0.0
  Change BL to M6 - Participant' acceptability for injection visits Q2M - Not at all acceptable | 1.1 | 1.6
  Change BL to M12 - Participant' acceptability for injection visits Q2M - Very acceptable: number analyzed (Participants) | 76 | 63
  Change BL to M12 - Participant' acceptability for injection visits Q2M - Very acceptable | -3.2 | -10.5
  Change BL to M12 - Participant' acceptability for injection visits Q2M - Acceptable: number analyzed (Participants) | 76 | 63
  Change BL to M12 - Participant' acceptability for injection visits Q2M - Acceptable | -1.9 | 3.6
  Change BL to M12 - Participant' acceptability for injection visits Q2M - Somewhat acceptable: number analyzed (Participants) | 76 | 63
  Change BL to M12 - Participant' acceptability for injection visits Q2M - Somewhat acceptable | 4.9 | 5.3
  Change BL to M12 - Participant' acceptability for injection visits Q2M - A little acceptable: number analyzed (Participants) | 76 | 63
  Change BL to M12 - Participant' acceptability for injection visits Q2M - A little acceptable | 0.1 | 1.6
  Change BL to M12 - Participant' acceptability for injection visits Q2M - Not at all acceptable: number analyzed (Participants) | 76 | 63
  Change BL to M12 - Participant' acceptability for injection visits Q2M - Not at all acceptable | 0.0 | 0.0

15. Secondary Outcome: Number of PSPs Assessed for Perception of Facilitators to Feasibility and Acceptability of APRETUDE Through Month 12
Description: Facilitators to feasibility and acceptability of APRETUDE measured from themes emerging from Proctor and Consolidated Framework for Implementation Research (CFIR) guided semi-structured qualitative interviews. In this outcome measure, PSPs were asked about their perception of the facilitators of feasibility and acceptability of APRETUDE intervention.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who completed an interview at the specified time point. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 23 | 21
Participants
  APRETUDE positive experience so far | 23 | 20
  Positive Experiences and General Satisfaction | 14 | 12
  Convenience and Ease of Use | 15 | 11
  Perceived effectiveness provides peace of mind | 7 | 2
  Discomfort becoming more manageable | 1 | 5
  APRETUDE met their expectations | 15 | 18
  Reduced anxiety about taking oral PrEP | 5 | 15
  HIV protection | 10 | 7
  APRETUDE more convenient than expected | 2 | 4

16. Secondary Outcome: Number of PSPs Assessed for Perception of Barriers to Feasibility and Acceptability of APRETUDE Through Month 12
Description: Barriers to feasibility and acceptability of APRETUDE were measured from themes emerging from Proctor and Consolidated Framework for Implementation Research (CFIR) guided semi-structured qualitative interviews. In this outcome measure, PSPs were asked about their perspectives on the barriers and challenges of feasibility and acceptability of APRETUDE intervention.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 23 | 21
Participants | 1 | 3

17. Secondary Outcome: Mean FIM Score for Telehealth Delivery Assessed for SSPs
Description: The FIM-TEL services for SSPs were a four-item measure (1. Telehealth for APRETUDE seems implementable in our clinic/practice 2. Telehealth for APRETUDE seems possible in our clinic/practice 3. Telehealth for APRETUDE seems doable in our clinic/practice 4. Telehealth for APRETUDE seems easy to use in our clinic/practice) and was measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least feasibility and 5 the most feasibility.
  Timeframe for evaluation of this outcome measure is BL, M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: At Baseline (Month 1), Month 4 and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 56 | 30
Scores on a scale
  Baseline | 4.01 (0.83) | 3.43 (1.23)
  Month 4: number analyzed (Participants) | 29 | 10
  Month 4 | 4.13 (0.90) | 4.08 (1.20)
  Month 12: number analyzed (Participants) | 30 | 9
  Month 12 | 4.26 (0.70) | 4.22 (1.30)

18. Secondary Outcome: Mean AIM Score for Telehealth Delivery Assessed for SSPs
Description: The AIM-TEL services for SSPs were a four-item measure (1. The idea of telehealth for APRETUDE in our clinic/practice meets my approval 2. The idea of telehealth for APRETUDE in our clinic/practice is appealing to me 3. I like the idea of telehealth for APRETUDE in our clinic/practice 4. I welcome the idea of telehealth for APRETUDE in our clinic/practice), each with a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least acceptability and 5 the most acceptability.
  Timeframe for evaluation of this outcome measure is BL, M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: At Baseline (Month 1), Month 4 and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 56 | 30
Scores on a scale
  Baseline | 4.09 (0.82) | 3.26 (1.38)
  Month 4: number analyzed (Participants) | 29 | 10
  Month 4 | 4.16 (0.78) | 3.98 (1.16)
  Month 12: number analyzed (Participants) | 30 | 9
  Month 12 | 4.07 (0.78) | 4.17 (1.28)

19. Secondary Outcome: Number of SSPs With Responses to the ISQs Regarding Use of Telehealth Delivery
Description: The ISQ used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, SSPs were asked about the use of telehealth services at their clinic/practice.
  Timeframe for evaluation of this outcome measure is BL, M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: At Baseline (Month 1), Month 4 and Month 12
Population: Analysis was performed on SSPs who completed at least one survey at any timepoint. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 56 | 30
Participants
  Month 1 - Does your clinic/practice use any form of telehealth for APRETUDE delivery?: Yes | 54 | 28
  Month 1 - Does your clinic/practice use any form of telehealth for APRETUDE delivery?: No | 1 | 0
  Month 1 - Does your clinic/practice use any form of telehealth for APRETUDE delivery?: I Don't Know | 1 | 2
  Month 4 - Does your clinic/practice use any form of telehealth for APRETUDE delivery?: number analyzed (Participants) | 51 | 29
  Month 4 - Does your clinic/practice use any form of telehealth for APRETUDE delivery?: Yes | 29 | 10
  Month 4 - Does your clinic/practice use any form of telehealth for APRETUDE delivery?: No | 15 | 14
  Month 4 - Does your clinic/practice use any form of telehealth for APRETUDE delivery?: I Don't Know | 7 | 5
  Month 12 - Does your clinic/practice use any form of telehealth for APRETUDE delivery?: number analyzed (Participants) | 52 | 29
  Month 12 - Does your clinic/practice use any form of telehealth for APRETUDE delivery?: Yes | 30 | 9
  Month 12 - Does your clinic/practice use any form of telehealth for APRETUDE delivery?: No | 11 | 12
  Month 12 - Does your clinic/practice use any form of telehealth for APRETUDE delivery?: I Don't Know | 11 | 8

20. Secondary Outcome: Number of SSPs With Responses to the ISQs Indicating Which Telehealth Services Were Used
Description: The ISQ used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, SSPs were asked about which telehealth services/systems were used at their clinic/practice to deliver APRETUDE during the PILLAR study.
  Timeframe for evaluation of this outcome measure is M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: At Month 4 and Month 12
Population: Analysis was performed on the SSPs who completed at least one survey at any time point. The use and adoption of these telehealth services were only assessed among DI SSPs at M4 but were assessed among both DI and RI SSPs at M12.
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 30 | 9
Participants
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: number analyzed (Participants) | 29 | 0
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: Yes, at my clinic's service/system | 14 | 0
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: Yes, services/systems offered through PILLAR study | 1 | 0
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: No | 8 | 0
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: I don't know | 6 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: number analyzed (Participants) | 29 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: Yes, at my clinic's service/system | 23 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: Yes, services/systems offered through PILLAR study | 1 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: No | 1 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: I don't know | 4 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: number analyzed (Participants) | 29 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: Yes, at my clinic's service/system | 4 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: Yes, services/systems offered through PILLAR study | 3 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: No | 17 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: I don't know | 5 | 0
  Month 4 - Injection appointment reminders: text/digital/email: number analyzed (Participants) | 29 | 0
  Month 4 - Injection appointment reminders: text/digital/email: Yes, at my clinic's service/system | 21 | 0
  Month 4 - Injection appointment reminders: text/digital/email: Yes, services/systems offered through PILLAR study | 1 | 0
  Month 4 - Injection appointment reminders: text/digital/email: No | 1 | 0
  Month 4 - Injection appointment reminders: text/digital/email: I don't know | 6 | 0
  Month 4 - HIV testing services: at home nurse testing: number analyzed (Participants) | 29 | 0
  Month 4 - HIV testing services: at home nurse testing: Yes, at my clinic's service/system | 8 | 0
  Month 4 - HIV testing services: at home nurse testing: Yes, services/systems offered through PILLAR study | 3 | 0
  Month 4 - HIV testing services: at home nurse testing: No | 14 | 0
  Month 4 - HIV testing services: at home nurse testing: I don't know | 4 | 0
  Month 12 - Online system for scheduling/rescheduling consultations and injection appointments: Yes, at my clinic's service/system | 21 | 5
  Month 12 - Online system for scheduling/rescheduling consultations and injection appointments: Yes, services/systems offered through PILLAR study | 1 | 1
  Month 12 - Online system for scheduling/rescheduling consultations and injection appointments: No | 5 | 3
  Month 12 - Online system for scheduling/rescheduling consultations and injection appointments: I don't know | 3 | 0
  Month 12 - Video/virtual consultations for initial and follow-up visits: Yes, at my clinic's service/system | 24 | 6
  Month 12 - Video/virtual consultations for initial and follow-up visits: Yes, services/systems offered through PILLAR study | 2 | 1
  Month 12 - Video/virtual consultations for initial and follow-up visits: No | 2 | 2
  Month 12 - Video/virtual consultations for initial and follow-up visits: I don't know | 2 | 0
  Month 12 - Injection Administration: home health nurse to administer injection: Yes, at my clinic's service/system | 6 | 1
  Month 12 - Injection Administration: home health nurse to administer injection: Yes, services/systems offered through PILLAR study | 6 | 1
  Month 12 - Injection Administration: home health nurse to administer injection: No | 16 | 7
  Month 12 - Injection Administration: home health nurse to administer injection: I don't know | 2 | 0
  Month 12 - Injection appointment reminders: text/digital/email: Yes, at my clinic's service/system | 23 | 5
  Month 12 - Injection appointment reminders: text/digital/email: Yes, services/systems offered through PILLAR study | 1 | 1
  Month 12 - Injection appointment reminders: text/digital/email: No | 2 | 3
  Month 12 - Injection appointment reminders: text/digital/email: I don't know | 4 | 0
  Month 12 - HIV testing services: at home nurse testing: Yes, at my clinic's service/system | 9 | 1
  Month 12 - HIV testing services: at home nurse testing: Yes, services/systems offered through PILLAR study | 6 | 1
  Month 12 - HIV testing services: at home nurse testing: No | 13 | 7
  Month 12 - HIV testing services: at home nurse testing: I don't know | 2 | 0

21. Secondary Outcome: Number of SSPs With Responses to the ISQs Indicating the Helpfulness of Telehealth Services Used
Description: The ISQ used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, SSPs were asked about the helpfulness of the telehealth services/systems used at their clinic/practice.
  Timeframe for evaluation of this outcome measure is M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: At Month 4 and Month 12
Population: Analysis was performed on SSPs who completed at least one survey at any timepoint. The use and adoption of these telehealth services were only assessed among DI SSPs at M4, but were assessed among both DI and RI SSPs at M12.
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 26 | 7
Participants
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: number analyzed (Participants) | 15 | 0
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: Very helpful | 10 | 0
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: Helpful | 3 | 0
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: Somewhat helpful | 1 | 0
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: A little helpful | 0 | 0
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: Not at all helpful | 0 | 0
  Month 4 - Online system for scheduling/rescheduling consultations and injection appointments: I have not personally used this | 1 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: number analyzed (Participants) | 24 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: Very helpful | 14 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: Helpful | 5 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: Somewhat helpful | 2 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: A little helpful | 0 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: Not at all helpful | 0 | 0
  Month 4 - Video/virtual consultations for initial and follow-up visits: I have not personally used this | 3 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: number analyzed (Participants) | 7 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: Very helpful | 2 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: Helpful | 2 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: Somewhat helpful | 1 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: A little helpful | 0 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: Not at all helpful | 0 | 0
  Month 4 - Injection Administration: home health nurse to administer injection: I have not personally used this | 2 | 0
  Month 4 - Injection appointment reminders: text/digital/email: number analyzed (Participants) | 22 | 0
  Month 4 - Injection appointment reminders: text/digital/email: Very helpful | 14 | 0
  Month 4 - Injection appointment reminders: text/digital/email: Helpful | 3 | 0
  Month 4 - Injection appointment reminders: text/digital/email: Somewhat helpful | 1 | 0
  Month 4 - Injection appointment reminders: text/digital/email: A little helpful | 0 | 0
  Month 4 - Injection appointment reminders: text/digital/email: Not at all helpful | 1 | 0
  Month 4 - Injection appointment reminders: text/digital/email: I have not personally used this | 3 | 0
  Month 4 - HIV testing services: at home nurse testing: number analyzed (Participants) | 11 | 0
  Month 4 - HIV testing services: at home nurse testing: Very helpful | 3 | 0
  Month 4 - HIV testing services: at home nurse testing: Helpful | 2 | 0
  Month 4 - HIV testing services: at home nurse testing: Somewhat helpful | 1 | 0
  Month 4 - HIV testing services: at home nurse testing: A little helpful | 0 | 0
  Month 4 - HIV testing services: at home nurse testing: Not at all helpful | 1 | 0
  Month 4 - HIV testing services: at home nurse testing: I have not personally used this | 4 | 0
  Month 12 - Online system for scheduling/rescheduling consultations and injection appointments: number analyzed (Participants) | 22 | 6
  Month 12 - Online system for scheduling/rescheduling consultations and injection appointments: Very helpful | 9 | 4
  Month 12 - Online system for scheduling/rescheduling consultations and injection appointments: Helpful | 7 | 2
  Month 12 - Online system for scheduling/rescheduling consultations and injection appointments: Somewhat helpful | 4 | 0
  Month 12 - Online system for scheduling/rescheduling consultations and injection appointments: A little helpful | 0 | 0
  Month 12 - Online system for scheduling/rescheduling consultations and injection appointments: Not at all helpful | 0 | 0
  Month 12 - Online system for scheduling/rescheduling consultations and injection appointments: I have not personally used this | 2 | 0
  Month 12 - Video/virtual consultations for initial and follow-up visits: Very helpful | 13 | 4
  Month 12 - Video/virtual consultations for initial and follow-up visits: Helpful | 6 | 1
  Month 12 - Video/virtual consultations for initial and follow-up visits: Somewhat helpful | 3 | 2
  Month 12 - Video/virtual consultations for initial and follow-up visits: A little helpful | 0 | 0
  Month 12 - Video/virtual consultations for initial and follow-up visits: Not at all helpful | 0 | 0
  Month 12 - Video/virtual consultations for initial and follow-up visits: I have not personally used this | 4 | 0
  Month 12 - Injection Administration: home health nurse to administer injection: number analyzed (Participants) | 12 | 2
  Month 12 - Injection Administration: home health nurse to administer injection: Very helpful | 5 | 1
  Month 12 - Injection Administration: home health nurse to administer injection: Helpful | 2 | 0
  Month 12 - Injection Administration: home health nurse to administer injection: Somewhat helpful | 1 | 0
  Month 12 - Injection Administration: home health nurse to administer injection: A little helpful | 0 | 0
  Month 12 - Injection Administration: home health nurse to administer injection: Not at all helpful | 0 | 0
  Month 12 - Injection Administration: home health nurse to administer injection: I have not personally used this | 4 | 1
  Month 12 - Injection appointment reminders: text/digital/email: number analyzed (Participants) | 24 | 6
  Month 12 - Injection appointment reminders: text/digital/email: Very helpful | 16 | 4
  Month 12 - Injection appointment reminders: text/digital/email: Helpful | 4 | 2
  Month 12 - Injection appointment reminders: text/digital/email: Somewhat helpful | 1 | 0
  Month 12 - Injection appointment reminders: text/digital/email: A little helpful | 1 | 0
  Month 12 - Injection appointment reminders: text/digital/email: Not at all helpful | 0 | 0
  Month 12 - Injection appointment reminders: text/digital/email: I have not personally used this | 2 | 0
  Month 12 - HIV testing services: at home nurse testing: number analyzed (Participants) | 15 | 2
  Month 12 - HIV testing services: at home nurse testing: Very helpful | 9 | 1
  Month 12 - HIV testing services: at home nurse testing: Helpful | 1 | 0
  Month 12 - HIV testing services: at home nurse testing: Somewhat helpful | 1 | 0
  Month 12 - HIV testing services: at home nurse testing: A little helpful | 0 | 0
  Month 12 - HIV testing services: at home nurse testing: Not at all helpful | 0 | 0
  Month 12 - HIV testing services: at home nurse testing: I have not personally used this | 4 | 1

22. Secondary Outcome: Change From Baseline in FIM Score for Telehealth Delivery Assessed for SSPs
Description: The FIM telehealth services for SSPs were a four-item measure (1. Telehealth for APRETUDE seems implementable in our clinic/practice 2. Telehealth for APRETUDE seems possible in our clinic/practice 3. Telehealth for APRETUDE seems doable in our clinic/practice 4. Telehealth for APRETUDE seems easy to use in our clinic/practice) and was measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least feasibility and 5 the most feasibility.
  Timeframe for evaluation of this outcome measure is M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI) compared to Baseline (BL).
Time Frame: At Month 4 and Month 12 compared to baseline (Month 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 28 | 10
Scores on a scale
  Month 4 compared to BL | -0.11 (1.21) | 0.20 (1.21)
  Month 12 compared to BL: number analyzed (Participants) | 26 | 8
  Month 12 compared to BL | -0.06 (1.03) | 0.16 (0.64)

23. Secondary Outcome: Change From Baseline in AIM Score for Telehealth Delivery Assessed for SSPs
Description: This outcome assesses the change in AIM telehealth services for SSPs over time. The AIM telehealth services for SSPs were a four-item measure (1. The idea of telehealth for APRETUDE in our clinic/practice meets my approval 2. The idea of telehealth for APRETUDE in our clinic/practice is appealing to me 3. I like the idea of telehealth for APRETUDE in our clinic/practice 4. I welcome the idea of telehealth for APRETUDE in our clinic/practice), each with a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least acceptability and 5 the most acceptability.
  Timeframe for evaluation of this outcome measure is M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI) compared to Baseline (BL).
Time Frame: At Month 4 and Month 12 compared to baseline (Month 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 28 | 10
Scores on a scale
  Month 4 compared to BL | -0.13 (0.92) | 0.53 (1.21)
  Month 12 compared to BL: number analyzed (Participants) | 26 | 8
  Month 12 compared to BL | -0.38 (0.97) | 0.41 (1.02)

24. Secondary Outcome: Percentage of SSPs With Change From Baseline in ISQ Responses for Telehealth Delivery
Description: The ISQ used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, SSPs were asked about the use of telehealth services at their clinic/practice.
  Timeframe for evaluation of this outcome measure is BL, M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI). The change from baseline is calculated as a difference of percentages resulted at each timepoint as following: M4 minus (-) BL, and M12-BL.
Time Frame: At Month 4 and Month 12 compared to Baseline (Month 1)
Population: as for outcome 19
Measure: Number; unit: Percentage of participants
Groups:
- DI- SSP: Staff at sites offering APRETUDE injection for pre- exposure prophylaxis (PrEP). SSPs had access to enhanced toolkits, a digital health implementation strategy and implementation facilitation for APRETUDE.
- RI- SSP: Staff at sites offering APRETUDE injection for PrEP. SSPs had access to standard toolkits for APRETUDE to use as needed.
Arm/Group | DI- SSP | RI- SSP
Number analyzed (Participants) | 52 | 29
Percentage of participants
  Change BL to M4 - Does your clinic/practice use any form of telehealth for APRETUDE delivery? - YES: number analyzed (Participants) | 51 | 29
  Change BL to M4 - Does your clinic/practice use any form of telehealth for APRETUDE delivery? - YES | -39.6 | -58.9
  Change BL to M4 - Does your clinic/practice use any form of telehealth for APRETUDE delivery? - NO: number analyzed (Participants) | 51 | 29
  Change BL to M4 - Does your clinic/practice use any form of telehealth for APRETUDE delivery? - NO | 27.6 | 48.3
  Change BL to M4-Does clinic/practice use any form of telehealth for APRETUDE delivery?-I DON'T KNOW: number analyzed (Participants) | 51 | 29
  Change BL to M4-Does clinic/practice use any form of telehealth for APRETUDE delivery?-I DON'T KNOW | 11.9 | 10.6
  Change BL to M12 - Does your clinic/practice use any form of telehealth for APRETUDE delivery? - YES | -38.7 | -62.3
  Change BL to M12 - Does your clinic/practice use any form of telehealth for APRETUDE delivery? - NO | 19.4 | 41.4
  Change BL to M12-Does clinic/practice use any form of telehealth for APRETUDE delivery?-I DON'T KNOW | 19.4 | 20.9

25. Secondary Outcome: Mean FIM Score for Telehealth Delivery Assessed for PSPs
Description: The FIM telehealth services for PSPs were a four-item measure (1. Using telehealth for APRETUDE services seems workable in my life 2. Using telehealth for APRETUDE services seems possible in my life 3. Using telehealth for APRETUDE services seems doable in my life 4. Using telehealth for APRETUDE services seems easy in my life) and was measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least feasibility and 5 the most feasibility.
  Timeframe for evaluation of this outcome measure is BL, M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Baseline (Month 1), Month 6 and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 105 | 76
Scores on a scale
  Baseline | 4.40 (0.72) | 4.15 (0.97)
  Month 6: number analyzed (Participants) | 40 | 24
  Month 6 | 4.56 (0.56) | 4.19 (0.76)
  Month 12: number analyzed (Participants) | 29 | 25
  Month 12 | 4.25 (0.89) | 4.38 (0.70)

26. Secondary Outcome: Mean AIM Score for Telehealth Delivery Assessed for PSPs
Description: The AIM Telehealth services for PSPs were a four-item measure (1. Using telehealth for APRETUDE services meets my approval 2. Using telehealth for APRETUDE services is appealing to me 3. I like telehealth for APRETUDE services 4. I welcome using telehealth for APRETUDE services), each with a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least acceptability and 5 the most acceptability.
  Timepoints during which this outcome measure was evaluated were BL, M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI)
Time Frame: At Baseline (Month 1), Month 6 and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 105 | 76
Scores on a scale
  Baseline | 4.32 (0.76) | 4.13 (0.91)
  Month 6: number analyzed (Participants) | 40 | 24
  Month 6 | 4.56 (0.57) | 4.25 (0.70)
  Month 12: number analyzed (Participants) | 29 | 25
  Month 12 | 4.21 (0.93) | 4.27 (0.67)

27. Secondary Outcome: Number of PSPs With Responses to the ISQs Regarding Telehealth Use for APRETUDE
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs were asked about the use of telehealth (TEL) services such as completing forms online, video chatting with their provider, getting reminders about their injection, or scheduling injection appointments online.
  Timeframe for evaluation of this outcome measure is BL, M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Baseline (Month 1), Month 6 and Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  Baseline- Have you used any of the telehealth care options that your clinic offers?: number analyzed (Participants) | 86 | 58
  Baseline- Have you used any of the telehealth care options that your clinic offers?: Yes | 72 | 48
  Baseline- Have you used any of the telehealth care options that your clinic offers?: No | 14 | 10
  Baseline- Have you used any of the telehealth care options that your clinic offers?: I don't know | 0 | 0
  Baseline- Have you used any of the telehealth care options that your clinic offers?: Missing | 0 | 0
  Month 6 - Have you used telehealth for any APRETUDE services in the last 6 months?: Yes | 41 | 24
  Month 6 - Have you used telehealth for any APRETUDE services in the last 6 months?: No | 49 | 34
  Month 6 - Have you used telehealth for any APRETUDE services in the last 6 months?: I don't know | 4 | 7
  Month 6 - Have you used telehealth for any APRETUDE services in the last 6 months?: Missing | 23 | 19
  Month 6- TEL services received: Doctor ordering HIV test at a lab near home to take the test: number analyzed (Participants) | 41 | 24
  Month 6- TEL services received: Doctor ordering HIV test at a lab near home to take the test: Yes | 17 | 9
  Month 6- TEL services received: Doctor ordering HIV test at a lab near home to take the test: No | 22 | 14
  Month 6- TEL services received: Doctor ordering HIV test at a lab near home to take the test: I don't know | 1 | 1
  Month 6- TEL services received: Doctor ordering HIV test at a lab near home to take the test: Missing | 1 | 0
  Month 6- TEL services received: Nurse coming home to give an HIV test: number analyzed (Participants) | 41 | 24
  Month 6- TEL services received: Nurse coming home to give an HIV test: Yes | 3 | 2
  Month 6- TEL services received: Nurse coming home to give an HIV test: No | 36 | 21
  Month 6- TEL services received: Nurse coming home to give an HIV test: I don't know | 1 | 1
  Month 6- TEL services received: Nurse coming home to give an HIV test: Missing | 1 | 0
  Month 6- TEL services received: Receiving reminders about scheduled injection appointment: number analyzed (Participants) | 41 | 24
  Month 6- TEL services received: Receiving reminders about scheduled injection appointment: Yes | 36 | 22
  Month 6- TEL services received: Receiving reminders about scheduled injection appointment: No | 4 | 1
  Month 6- TEL services received: Receiving reminders about scheduled injection appointment: I don't know | 0 | 1
  Month 6- TEL services received: Receiving reminders about scheduled injection appointment: Missing | 1 | 0
  Month 6- TEL services received: Scheduling injection appointment online: number analyzed (Participants) | 41 | 24
  Month 6- TEL services received: Scheduling injection appointment online: Yes | 24 | 15
  Month 6- TEL services received: Scheduling injection appointment online: No | 15 | 8
  Month 6- TEL services received: Scheduling injection appointment online: I don't know | 1 | 1
  Month 6- TEL services received: Scheduling injection appointment online: Missing | 1 | 0
  Month 6- TEL services received: Nurse coming home to give the injection: number analyzed (Participants) | 41 | 24
  Month 6- TEL services received: Nurse coming home to give the injection: Yes | 2 | 2
  Month 6- TEL services received: Nurse coming home to give the injection: No | 38 | 21
  Month 6- TEL services received: Nurse coming home to give the injection: I don't know | 0 | 1
  Month 6- TEL services received: Nurse coming home to give the injection: Missing | 1 | 0
  Month 12 - Have you used telehealth for any APRETUDE services in the last 6 months?: Yes | 29 | 25
  Month 12 - Have you used telehealth for any APRETUDE services in the last 6 months?: No | 47 | 38
  Month 12 - Have you used telehealth for any APRETUDE services in the last 6 months?: I don't know | 1 | 0
  Month 12 - Have you used telehealth for any APRETUDE services in the last 6 months?: Missing | 40 | 21
  Month 12- TEL services received: Doctor ordering HIV test at a lab near home to take the test: number analyzed (Participants) | 29 | 25
  Month 12- TEL services received: Doctor ordering HIV test at a lab near home to take the test: Yes | 11 | 10
  Month 12- TEL services received: Doctor ordering HIV test at a lab near home to take the test: No | 17 | 13
  Month 12- TEL services received: Doctor ordering HIV test at a lab near home to take the test: I don't know | 1 | 2
  Month 12- TEL services received: Doctor ordering HIV test at a lab near home to take the test: Missing | 0 | 0
  Month 12- TEL services received: Nurse coming home to give an HIV test: number analyzed (Participants) | 29 | 25
  Month 12- TEL services received: Nurse coming home to give an HIV test: Yes | 3 | 2
  Month 12- TEL services received: Nurse coming home to give an HIV test: No | 26 | 23
  Month 12- TEL services received: Nurse coming home to give an HIV test: I don't know | 0 | 0
  Month 12- TEL services received: Nurse coming home to give an HIV test: Missing | 0 | 0
  Month 12- TEL services received: Receiving reminders about scheduled injection appointment: number analyzed (Participants) | 29 | 25
  Month 12- TEL services received: Receiving reminders about scheduled injection appointment: Yes | 28 | 25
  Month 12- TEL services received: Receiving reminders about scheduled injection appointment: No | 1 | 0
  Month 12- TEL services received: Receiving reminders about scheduled injection appointment: I don't know | 0 | 0
  Month 12- TEL services received: Receiving reminders about scheduled injection appointment: Missing | 0 | 0
  Month 12- TEL services received: Scheduling injection appointment online: number analyzed (Participants) | 29 | 25
  Month 12- TEL services received: Scheduling injection appointment online: Yes | 16 | 13
  Month 12- TEL services received: Scheduling injection appointment online: No | 13 | 12
  Month 12- TEL services received: Scheduling injection appointment online: I don't know | 0 | 0
  Month 12- TEL services received: Scheduling injection appointment online: Missing | 0 | 0
  Month 12- TEL services received: Nurse coming home to give the injection: number analyzed (Participants) | 29 | 25
  Month 12- TEL services received: Nurse coming home to give the injection: Yes | 3 | 2
  Month 12- TEL services received: Nurse coming home to give the injection: No | 25 | 23
  Month 12- TEL services received: Nurse coming home to give the injection: I don't know | 1 | 0
  Month 12- TEL services received: Nurse coming home to give the injection: Missing | 0 | 0

28. Secondary Outcome: Number of PSPs With Responses to the ISQs Regarding the Comfort of Using Telehealth Services
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs were asked about how comfortable it was to use various telehealth services for APRETUDE.
  Timeframe for evaluation of this outcome measure is M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Month 6 and Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 36 | 25
Participants
  Month 6- Doctor ordering HIV test at a lab near home to take the test: number analyzed (Participants) | 17 | 9
  Month 6- Doctor ordering HIV test at a lab near home to take the test: Very comfortable | 12 | 8
  Month 6- Doctor ordering HIV test at a lab near home to take the test: Somewhat comfortable | 4 | 1
  Month 6- Doctor ordering HIV test at a lab near home to take the test: Neither comfortable nor uncomfortable | 1 | 0
  Month 6- Doctor ordering HIV test at a lab near home to take the test: Somewhat uncomfortable | 0 | 0
  Month 6- Doctor ordering HIV test at a lab near home to take the test: Not comfortable at all | 0 | 0
  Month 6- A nurse coming home to give an HIV test: number analyzed (Participants) | 3 | 2
  Month 6- A nurse coming home to give an HIV test: Very comfortable | 2 | 1
  Month 6- A nurse coming home to give an HIV test: Somewhat comfortable | 0 | 1
  Month 6- A nurse coming home to give an HIV test: Neither comfortable nor uncomfortable | 1 | 0
  Month 6- A nurse coming home to give an HIV test: Somewhat uncomfortable | 0 | 0
  Month 6- A nurse coming home to give an HIV test: Not comfortable at all | 0 | 0
  Month 6- Receiving reminders about scheduled injection appointment: number analyzed (Participants) | 36 | 22
  Month 6- Receiving reminders about scheduled injection appointment: Very comfortable | 33 | 20
  Month 6- Receiving reminders about scheduled injection appointment: Somewhat comfortable | 3 | 2
  Month 6- Receiving reminders about scheduled injection appointment: Neither comfortable nor uncomfortable | 0 | 0
  Month 6- Receiving reminders about scheduled injection appointment: Somewhat uncomfortable | 0 | 0
  Month 6- Receiving reminders about scheduled injection appointment: Not comfortable at all | 0 | 0
  Month 6- Scheduling injection appointment online: number analyzed (Participants) | 24 | 15
  Month 6- Scheduling injection appointment online: Very comfortable | 20 | 13
  Month 6- Scheduling injection appointment online: Somewhat comfortable | 3 | 1
  Month 6- Scheduling injection appointment online: Neither comfortable nor uncomfortable | 0 | 1
  Month 6- Scheduling injection appointment online: Somewhat uncomfortable | 1 | 0
  Month 6- Scheduling injection appointment online: Not comfortable at all | 0 | 0
  Month 6- A nurse coming home to give the injection: number analyzed (Participants) | 2 | 2
  Month 6- A nurse coming home to give the injection: Very comfortable | 2 | 1
  Month 6- A nurse coming home to give the injection: Somewhat comfortable | 0 | 0
  Month 6- A nurse coming home to give the injection: Neither comfortable nor uncomfortable | 0 | 0
  Month 6- A nurse coming home to give the injection: Somewhat uncomfortable | 0 | 1
  Month 6- A nurse coming home to give the injection: Not comfortable at all | 0 | 0
  Month 12- Doctor ordering HIV test at a lab near home to take the test: number analyzed (Participants) | 11 | 10
  Month 12- Doctor ordering HIV test at a lab near home to take the test: Very comfortable | 11 | 8
  Month 12- Doctor ordering HIV test at a lab near home to take the test: Somewhat comfortable | 0 | 0
  Month 12- Doctor ordering HIV test at a lab near home to take the test: Neither comfortable nor uncomfortable | 0 | 2
  Month 12- Doctor ordering HIV test at a lab near home to take the test: Somewhat uncomfortable | 0 | 0
  Month 12- Doctor ordering HIV test at a lab near home to take the test: Not comfortable at all | 0 | 0
  Month 12- A nurse coming to home to give an HIV test: number analyzed (Participants) | 3 | 2
  Month 12- A nurse coming to home to give an HIV test: Very comfortable | 2 | 2
  Month 12- A nurse coming to home to give an HIV test: Somewhat comfortable | 1 | 0
  Month 12- A nurse coming to home to give an HIV test: Neither comfortable nor uncomfortable | 0 | 0
  Month 12- A nurse coming to home to give an HIV test: Somewhat uncomfortable | 0 | 0
  Month 12- A nurse coming to home to give an HIV test: Not comfortable at all | 0 | 0
  Month 12- Receiving reminders about scheduled injection appointment: number analyzed (Participants) | 28 | 25
  Month 12- Receiving reminders about scheduled injection appointment: Very comfortable | 26 | 21
  Month 12- Receiving reminders about scheduled injection appointment: Somewhat comfortable | 2 | 2
  Month 12- Receiving reminders about scheduled injection appointment: Neither comfortable nor uncomfortable | 0 | 1
  Month 12- Receiving reminders about scheduled injection appointment: Somewhat uncomfortable | 0 | 1
  Month 12- Receiving reminders about scheduled injection appointment: Not comfortable at all | 0 | 0
  Month 12- Scheduling injection appointment online: number analyzed (Participants) | 16 | 13
  Month 12- Scheduling injection appointment online: Very comfortable | 15 | 11
  Month 12- Scheduling injection appointment online: Somewhat comfortable | 1 | 1
  Month 12- Scheduling injection appointment online: Neither comfortable nor uncomfortable | 0 | 1
  Month 12- Scheduling injection appointment online: Somewhat uncomfortable | 0 | 0
  Month 12- Scheduling injection appointment online: Not comfortable at all | 0 | 0
  Month 12- A nurse coming home to give the injection: number analyzed (Participants) | 3 | 2
  Month 12- A nurse coming home to give the injection: Very comfortable | 3 | 2
  Month 12- A nurse coming home to give the injection: Somewhat comfortable | 0 | 0
  Month 12- A nurse coming home to give the injection: Neither comfortable nor uncomfortable | 0 | 0
  Month 12- A nurse coming home to give the injection: Somewhat uncomfortable | 0 | 0
  Month 12- A nurse coming home to give the injection: Not comfortable at all | 0 | 0

29. Secondary Outcome: Number of PSPs With Response to the ISQs Regarding the Convenience of Telehealth Services Used
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs were asked about how convenient it was to use various telehealth services for APRETUDE.
  Timeframe for evaluation of this outcome measure is M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Month 6 and Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 36 | 25
Participants
  Month 6- Doctor ordering HIV test at a lab near home to take the test: number analyzed (Participants) | 17 | 9
  Month 6- Doctor ordering HIV test at a lab near home to take the test: Very convenient | 12 | 8
  Month 6- Doctor ordering HIV test at a lab near home to take the test: Somewhat convenient | 3 | 0
  Month 6- Doctor ordering HIV test at a lab near home to take the test: Neither convenient nor inconvenient | 2 | 1
  Month 6- Doctor ordering HIV test at a lab near home to take the test: Somewhat inconvenient | 0 | 0
  Month 6- Doctor ordering HIV test at a lab near home to take the test: Very inconvenient | 0 | 0
  Month 6- A nurse coming home to give an HIV test: number analyzed (Participants) | 3 | 2
  Month 6- A nurse coming home to give an HIV test: Very convenient | 1 | 2
  Month 6- A nurse coming home to give an HIV test: Somewhat convenient | 1 | 0
  Month 6- A nurse coming home to give an HIV test: Neither convenient nor inconvenient | 1 | 0
  Month 6- A nurse coming home to give an HIV test: Somewhat inconvenient | 0 | 0
  Month 6- A nurse coming home to give an HIV test: Very inconvenient | 0 | 0
  Month 6- Receiving reminders about scheduled injection appointment: number analyzed (Participants) | 36 | 22
  Month 6- Receiving reminders about scheduled injection appointment: Very convenient | 31 | 18
  Month 6- Receiving reminders about scheduled injection appointment: Somewhat convenient | 4 | 4
  Month 6- Receiving reminders about scheduled injection appointment: Neither convenient nor inconvenient | 1 | 0
  Month 6- Receiving reminders about scheduled injection appointment: Somewhat inconvenient | 0 | 0
  Month 6- Receiving reminders about scheduled injection appointment: Very inconvenient | 0 | 0
  Month 6- Scheduling your injection appointment online: number analyzed (Participants) | 24 | 15
  Month 6- Scheduling your injection appointment online: Very convenient | 19 | 13
  Month 6- Scheduling your injection appointment online: Somewhat convenient | 3 | 1
  Month 6- Scheduling your injection appointment online: Neither convenient nor inconvenient | 2 | 0
  Month 6- Scheduling your injection appointment online: Somewhat inconvenient | 0 | 1
  Month 6- Scheduling your injection appointment online: Very inconvenient | 0 | 0
  Month 6- A nurse coming home to give the injection: number analyzed (Participants) | 2 | 2
  Month 6- A nurse coming home to give the injection: Very convenient | 2 | 1
  Month 6- A nurse coming home to give the injection: Somewhat convenient | 0 | 0
  Month 6- A nurse coming home to give the injection: Neither convenient nor inconvenient | 0 | 0
  Month 6- A nurse coming home to give the injection: Somewhat inconvenient | 0 | 0
  Month 6- A nurse coming home to give the injection: Very inconvenient | 0 | 1
  Month 12- Doctor ordering HIV test at a lab near home to take the test: number analyzed (Participants) | 11 | 10
  Month 12- Doctor ordering HIV test at a lab near home to take the test: Very convenient | 11 | 9
  Month 12- Doctor ordering HIV test at a lab near home to take the test: Somewhat convenient | 0 | 0
  Month 12- Doctor ordering HIV test at a lab near home to take the test: Neither convenient nor inconvenient | 0 | 1
  Month 12- Doctor ordering HIV test at a lab near home to take the test: Somewhat inconvenient | 0 | 0
  Month 12- Doctor ordering HIV test at a lab near home to take the test: Very inconvenient | 0 | 0
  Month 12- A nurse coming home to give an HIV test: number analyzed (Participants) | 3 | 2
  Month 12- A nurse coming home to give an HIV test: Very convenient | 2 | 2
  Month 12- A nurse coming home to give an HIV test: Somewhat convenient | 1 | 0
  Month 12- A nurse coming home to give an HIV test: Neither convenient nor inconvenient | 0 | 0
  Month 12- A nurse coming home to give an HIV test: Somewhat inconvenient | 0 | 0
  Month 12- A nurse coming home to give an HIV test: Very inconvenient | 0 | 0
  Month 12- Receiving reminders about scheduled injection appointment: number analyzed (Participants) | 28 | 25
  Month 12- Receiving reminders about scheduled injection appointment: Very convenient | 28 | 22
  Month 12- Receiving reminders about scheduled injection appointment: Somewhat convenient | 0 | 2
  Month 12- Receiving reminders about scheduled injection appointment: Neither convenient nor inconvenient | 0 | 1
  Month 12- Receiving reminders about scheduled injection appointment: Somewhat inconvenient | 0 | 0
  Month 12- Receiving reminders about scheduled injection appointment: Very inconvenient | 0 | 0
  Month 12- Scheduling your injection appointment online: number analyzed (Participants) | 16 | 13
  Month 12- Scheduling your injection appointment online: Very convenient | 14 | 11
  Month 12- Scheduling your injection appointment online: Somewhat convenient | 1 | 1
  Month 12- Scheduling your injection appointment online: Neither convenient nor inconvenient | 1 | 1
  Month 12- Scheduling your injection appointment online: Somewhat inconvenient | 0 | 0
  Month 12- Scheduling your injection appointment online: Very inconvenient | 0 | 0
  Month 12- A nurse coming home to give the injection: number analyzed (Participants) | 3 | 2
  Month 12- A nurse coming home to give the injection: Very convenient | 3 | 2
  Month 12- A nurse coming home to give the injection: Somewhat convenient | 0 | 0
  Month 12- A nurse coming home to give the injection: Neither convenient nor inconvenient | 0 | 0
  Month 12- A nurse coming home to give the injection: Somewhat inconvenient | 0 | 0
  Month 12- A nurse coming home to give the injection: Very inconvenient | 0 | 0

30. Secondary Outcome: Number of PSPs With Response to the ISQs Recommending Telehealth Delivery
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs were asked if they would recommend telehealth services for APRETUDE to other people.
  Timeframe for evaluation of this outcome measure is M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI).
Time Frame: At Month 6 and Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 41 | 25
Participants
  Month 6 - I would recommend telehealth services for APRETUDE to other people.: number analyzed (Participants) | 41 | 24
  Month 6 - I would recommend telehealth services for APRETUDE to other people.: Completely agree | 29 | 12
  Month 6 - I would recommend telehealth services for APRETUDE to other people.: Agree | 9 | 9
  Month 6 - I would recommend telehealth services for APRETUDE to other people.: Neither agree not disagree | 1 | 3
  Month 6 - I would recommend telehealth services for APRETUDE to other people.: Disagree | 1 | 0
  Month 6 - I would recommend telehealth services for APRETUDE to other people.: Completely disagree | 0 | 0
  Month 6 - I would recommend telehealth services for APRETUDE to other people.: Missing | 1 | 0
  Month 12 - I would recommend telehealth services for APRETUDE to other people.: number analyzed (Participants) | 29 | 25
  Month 12 - I would recommend telehealth services for APRETUDE to other people.: Completely agree | 20 | 20
  Month 12 - I would recommend telehealth services for APRETUDE to other people.: Agree | 7 | 2
  Month 12 - I would recommend telehealth services for APRETUDE to other people.: Neither agree not disagree | 2 | 3
  Month 12 - I would recommend telehealth services for APRETUDE to other people.: Disagree | 0 | 0
  Month 12 - I would recommend telehealth services for APRETUDE to other people.: Completely disagree | 0 | 0
  Month 12 - I would recommend telehealth services for APRETUDE to other people.: Missing | 0 | 0

31. Secondary Outcome: Change From Baseline in FIM Score for Telehealth Delivery Assessed for PSPs
Description: The FIM Telehealth services for PSPs were a four-item measure (1. Using telehealth for APRETUDE services seems workable in my life 2. Using telehealth for APRETUDE services seems possible in my life 3. Using telehealth for APRETUDE services seems doable in my life 4. Using telehealth for APRETUDE services seems easy in my life) and was measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least feasibility and 5 the most feasibility.
  Timeframe for evaluation of this outcome measure is M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI) compared to BL.
Time Frame: At Month 6 and Month 12 compared to baseline (Month 1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 37 | 23
Scores on a scale
  Month 6 compared to BL: number analyzed (Participants) | 37 | 22
  Month 6 compared to BL | 0.08 (0.65) | 0.25 (1.23)
  Month 12 compared to BL: number analyzed (Participants) | 27 | 23
  Month 12 compared to BL | -0.35 (0.78) | 0.17 (1.21)

32. Secondary Outcome: Change From Baseline in AIM Score for Telehealth Delivery Assessed for PSPs
Description: The AIM Telehealth services for PSPs were a four-item measure (1. Using telehealth for APRETUDE services meets my approval 2. Using telehealth for APRETUDE services is appealing to me 3. I like telehealth for APRETUDE services 4. I welcome using telehealth for APRETUDE services), each with a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least acceptability and 5 the most acceptability.
  Timeframe for evaluation of this outcome measure is M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI) compared to BL.
Time Frame: At Month 6 and Month 12 compared to baseline (Month 1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 37 | 23
Scores on a scale
  Month 6 compared to BL: number analyzed (Participants) | 37 | 22
  Month 6 compared to BL | 0.09 (0.64) | 0.26 (1.26)
  Month 12 compared to BL: number analyzed (Participants) | 27 | 23
  Month 12 compared to BL | -0.39 (0.92) | 0.21 (1.11)

33. Secondary Outcome: Percentage of PSPs With Change From Baseline in ISQ Responses Regarding Telehealth Delivery
Description: The ISQ used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs were asked about the use of telehealth (TEL) services such as completing forms online, video chatting with their provider, getting reminders about their injection, or scheduling injection appointments online.
  Timeframe for evaluation of this outcome measure is BL, M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI). The change from baseline is calculated as a difference of percentages resulted at each timepoint as following: M6 minus (-) BL, and M12-BL.
Time Frame: At Month 6 and Month 12 compared to Baseline (Month 1)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | DI- PSP | RI- PSP
Number analyzed (Participants) | 94 | 65
Percentage of participants
  Change BL to M6-Have you used telehealth for any APRETUDE services in the last 6 months? - YES | -40.1 | -45.8
  Change BL to M6-Have you used telehealth for any APRETUDE services in the last 6 months? - NO | 35.8 | 35.1
  Change BL to M6-Have you used telehealth for any APRETUDE services in the last 6 months?-DON'T KNOW | 4.3 | 10.8
  Change BL to M12 - Have you used telehealth for any APRETUDE services in the last 6 months? - YES: number analyzed (Participants) | 77 | 63
  Change BL to M12 - Have you used telehealth for any APRETUDE services in the last 6 months? - YES | -46.1 | -43.1
  Change BL to M12 - Have you used telehealth for any APRETUDE services in the last 6 months? - NO: number analyzed (Participants) | 77 | 63
  Change BL to M12 - Have you used telehealth for any APRETUDE services in the last 6 months? - NO | 44.8 | 43.1
  Change BL to M12-Have you used telehealth for any APRETUDE services in the last 6 months?-DON'T KNOW: number analyzed (Participants) | 77 | 63
  Change BL to M12-Have you used telehealth for any APRETUDE services in the last 6 months?-DON'T KNOW | 1.3 | 0.0

34. Secondary Outcome: Number of SSPs Assessed for Perception of Facilitators and Barriers to Feasibility and Acceptability for Telehealth Delivery
Description: Barriers and facilitators to the feasibility and acceptability of telehealth use for APRETUDE were measured from themes emerging from Proctor and Consolidated Framework for Implementation Research (CFIR) guided semi-structured qualitative interviews. In this outcome measure, SSPs were asked their perceptions of these facilitators and barriers for telehealth services used.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 27 | 8
Participants
  Video consultation: Very easy | 12 | 4
  Video consultation: Somewhat easy | 3 | 2
  Video consultation: Neither easy nor difficult | 6 | 1
  Video consultation: Somewhat Difficult | 0 | 0
  Video consultation: Very Difficult | 0 | 0
  Video consultation: I don't use this system | 6 | 1
  Telephone consultation: number analyzed (Participants) | 25 | 4
  Telephone consultation: Very easy | 14 | 2
  Telephone consultation: Somewhat easy | 4 | 2
  Telephone consultation: Neither easy nor difficult | 3 | 0
  Telephone consultation: Somewhat Difficult | 1 | 0
  Telephone consultation: Very Difficult | 0 | 0
  Telephone consultation: I don't use this system | 3 | 0
  Remote monitoring of patients: number analyzed (Participants) | 11 | 3
  Remote monitoring of patients: Very easy | 3 | 1
  Remote monitoring of patients: Somewhat easy | 5 | 0
  Remote monitoring of patients: Neither easy nor difficult | 2 | 1
  Remote monitoring of patients: Somewhat Difficult | 0 | 0
  Remote monitoring of patients: Very Difficult | 0 | 0
  Remote monitoring of patients: I don't use this system | 1 | 1
  Online appointment scheduling: number analyzed (Participants) | 10 | 3
  Online appointment scheduling: Very easy | 3 | 3
  Online appointment scheduling: Somewhat easy | 2 | 0
  Online appointment scheduling: Neither easy nor difficult | 3 | 0
  Online appointment scheduling: Somewhat Difficult | 0 | 0
  Online appointment scheduling: Very Difficult | 0 | 0
  Online appointment scheduling: I don't use this system | 2 | 0
  Patient portal conversations: ability for patients to send messages to providers: number analyzed (Participants) | 23 | 8
  Patient portal conversations: ability for patients to send messages to providers: Very easy | 13 | 7
  Patient portal conversations: ability for patients to send messages to providers: Somewhat easy | 4 | 0
  Patient portal conversations: ability for patients to send messages to providers: Neither easy nor difficult | 4 | 0
  Patient portal conversations: ability for patients to send messages to providers: Somewhat Difficult | 0 | 1
  Patient portal conversations: ability for patients to send messages to providers: Very Difficult | 0 | 0
  Patient portal conversations: ability for patients to send messages to providers: I don't use this system | 2 | 0
  At-home testing services: number analyzed (Participants) | 10 | 2
  At-home testing services: Very easy | 4 | 1
  At-home testing services: Somewhat easy | 1 | 1
  At-home testing services: Neither easy nor difficult | 2 | 0
  At-home testing services: Somewhat Difficult | 0 | 0
  At-home testing services: Very Difficult | 0 | 0
  At-home testing services: I don't use this system | 3 | 0
  Send and receiving patient reported outcomes questionnaires via an online system: number analyzed (Participants) | 12 | 2
  Send and receiving patient reported outcomes questionnaires via an online system: Very easy | 3 | 1
  Send and receiving patient reported outcomes questionnaires via an online system: Somewhat easy | 4 | 1
  Send and receiving patient reported outcomes questionnaires via an online system: Neither easy nor difficult | 3 | 0
  Send and receiving patient reported outcomes questionnaires via an online system: Somewhat Difficult | 0 | 0
  Send and receiving patient reported outcomes questionnaires via an online system: Very Difficult | 0 | 0
  Send and receiving patient reported outcomes questionnaires via an online system: I don't use this system | 2 | 0
  Online prescription refills: number analyzed (Participants) | 23 | 6
  Online prescription refills: Very easy | 14 | 6
  Online prescription refills: Somewhat easy | 3 | 0
  Online prescription refills: Neither easy nor difficult | 4 | 0
  Online prescription refills: Somewhat Difficult | 0 | 0
  Online prescription refills: Very Difficult | 0 | 0
  Online prescription refills: I don't use this system | 2 | 0
  Online portal for patients to access medical documents, such as visit summaries and test results: number analyzed (Participants) | 24 | 6
  Online portal for patients to access medical documents, such as visit summaries and test results: Very easy | 12 | 6
  Online portal for patients to access medical documents, such as visit summaries and test results: Somewhat easy | 6 | 0
  Online portal for patients to access medical documents, such as visit summaries and test results: Neither easy nor difficult | 4 | 0
  Online portal for patients to access medical documents, such as visit summaries and test results: Somewhat Difficult | 0 | 0
  Online portal for patients to access medical documents, such as visit summaries and test results: Very Difficult | 0 | 0
  Online portal for patients to access medical documents, such as visit summaries and test results: I don't use this system | 2 | 0
  Text messaging with patients about care: number analyzed (Participants) | 13 | 6
  Text messaging with patients about care: Very easy | 7 | 4
  Text messaging with patients about care: Somewhat easy | 3 | 1
  Text messaging with patients about care: Neither easy nor difficult | 2 | 1
  Text messaging with patients about care: Somewhat Difficult | 0 | 0
  Text messaging with patients about care: Very Difficult | 0 | 0
  Text messaging with patients about care: I don't use this system | 1 | 0
  Email reminders to patient about upcoming visits: number analyzed (Participants) | 19 | 4
  Email reminders to patient about upcoming visits: Very easy | 10 | 3
  Email reminders to patient about upcoming visits: Somewhat easy | 4 | 1
  Email reminders to patient about upcoming visits: Neither easy nor difficult | 2 | 0
  Email reminders to patient about upcoming visits: Somewhat Difficult | 0 | 0
  Email reminders to patient about upcoming visits: Very Difficult | 0 | 0
  Email reminders to patient about upcoming visits: I don't use this system | 3 | 0
  Text reminders: number analyzed (Participants) | 22 | 8
  Text reminders: Very easy | 12 | 6
  Text reminders: Somewhat easy | 5 | 1
  Text reminders: Neither easy nor difficult | 2 | 1
  Text reminders: Somewhat Difficult | 0 | 0
  Text reminders: Very Difficult | 0 | 0
  Text reminders: I don't use this system | 3 | 0
  Automated phone call reminders: number analyzed (Participants) | 19 | 5
  Automated phone call reminders: Very easy | 9 | 4
  Automated phone call reminders: Somewhat easy | 4 | 1
  Automated phone call reminders: Neither easy nor difficult | 4 | 0
  Automated phone call reminders: Somewhat Difficult | 0 | 0
  Automated phone call reminders: Very Difficult | 0 | 0
  Automated phone call reminders: I don't use this system | 2 | 0
  Staff phone call reminder: number analyzed (Participants) | 18 | 8
  Staff phone call reminder: Very easy | 9 | 7
  Staff phone call reminder: Somewhat easy | 6 | 1
  Staff phone call reminder: Neither easy nor difficult | 1 | 0
  Staff phone call reminder: Somewhat Difficult | 0 | 0
  Staff phone call reminder: Very Difficult | 0 | 0
  Staff phone call reminder: I don't use this system | 2 | 0
  Sending motivational reminders to help patients persist on APRETUDE: number analyzed (Participants) | 2 | 1
  Sending motivational reminders to help patients persist on APRETUDE: Very easy | 2 | 1
  Sending motivational reminders to help patients persist on APRETUDE: Somewhat easy | 0 | 0
  Sending motivational reminders to help patients persist on APRETUDE: Neither easy nor difficult | 0 | 0
  Sending motivational reminders to help patients persist on APRETUDE: Somewhat Difficult | 0 | 0
  Sending motivational reminders to help patients persist on APRETUDE: Very Difficult | 0 | 0
  Sending motivational reminders to help patients persist on APRETUDE: I don't use this system | 0 | 0
  Sending cabotegravir oral lead in to patient's home: number analyzed (Participants) | 7 | 2
  Sending cabotegravir oral lead in to patient's home: Very easy | 4 | 1
  Sending cabotegravir oral lead in to patient's home: Somewhat easy | 1 | 0
  Sending cabotegravir oral lead in to patient's home: Neither easy nor difficult | 1 | 1
  Sending cabotegravir oral lead in to patient's home: Somewhat Difficult | 0 | 0
  Sending cabotegravir oral lead in to patient's home: Very Difficult | 0 | 0
  Sending cabotegravir oral lead in to patient's home: I don't use this system | 1 | 0
  Insurance/benefits verification: number analyzed (Participants) | 24 | 7
  Insurance/benefits verification: Very easy | 10 | 5
  Insurance/benefits verification: Somewhat easy | 7 | 1
  Insurance/benefits verification: Neither easy nor difficult | 3 | 1
  Insurance/benefits verification: Somewhat Difficult | 1 | 0
  Insurance/benefits verification: Very Difficult | 1 | 0
  Insurance/benefits verification: I don't use this system | 2 | 0

35. Secondary Outcome: Number of PSPs Assessed for Perception of Facilitators and Barriers to Feasibility and Acceptability for Telehealth Delivery
Description: Barriers and facilitators to the feasibility and acceptability of telehealth use for APRETUDE were measured from themes emerging from Proctor and Consolidated Framework for Implementation Research (CFIR) guided semi-structured qualitative interviews. In this outcome measure, PSPs were asked their perceptions of these facilitators and barriers for telehealth services used.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who completed an interview at the specified time point. The use and adoption of some telehealth services were only assessed among DI PSPs. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 23 | 21
Participants
  Telehealth Used for any service | 2 | 5
  Telehealth Used for APRETUDE | 1 | 5
  Telehealth used for things OTHER than APRETUDE, only | 1 | 0
  Telehealth Not Used | 2 | 12
  Not Asked About Telehealth | 18 | 4
  Telehealth used/not used- Missing | 1 | 0
  Telehealth DI Used: number analyzed (Participants) | 17 | 0
  Telehealth DI Used | 5 | 0
  Teleconsultant Used: number analyzed (Participants) | 17 | 0
  Teleconsultant Used | 1 | 0
  Online Appointment Scheduler Used: number analyzed (Participants) | 17 | 0
  Online Appointment Scheduler Used | 0 | 0
  Reminders Used: number analyzed (Participants) | 17 | 0
  Reminders Used | 3 | 0
  Home tests Used: number analyzed (Participants) | 17 | 0
  Home tests Used | 0 | 0
  Local labs Used: number analyzed (Participants) | 17 | 0
  Local labs Used | 0 | 0
  Online portal Used: number analyzed (Participants) | 17 | 0
  Online portal Used | 0 | 0
  Home health nurses Used: number analyzed (Participants) | 17 | 0
  Home health nurses Used | 0 | 0
  Screenings and assessments Used: number analyzed (Participants) | 17 | 0
  Screenings and assessments Used | 1 | 0

36. Secondary Outcome: Mean AIM Score Assessed for SSPs
Description: AIM score for SSPs has 2 parts- AIM-INT that evaluates perceived intervention acceptability among SSPs and consists of 4 items (1. APRETUDE in our clinic/practice meets my approval 2. APRETUDE in our clinic/practice is appealing to me 3. I like APRETUDE in our clinic/practice 4. I welcome APRETUDE in our clinic/practice), and AIM-Implementation (IMP) that evaluates perceived acceptability of DI and RI approaches among SSPs and consists of 4 items (1. The implementation support has met my approval; 2. The implementation support was appealing to me; 3. I like the implementation support I have received; 4. I welcome the implementation support I have received),each with a five-point rating scale (1=completely disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, and 5=completely agree). Mean score ranges from 1 to 5 with 1=least acceptability and 5=most acceptability.
  Timeframe for evaluation is BL, M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: At Baseline (Month 1), Month 4 and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 56 | 30
Scores on a scale
  AIM-INT (Baseline) | 4.69 (0.43) | 4.66 (0.48)
  AIM-INT (Month 4): number analyzed (Participants) | 51 | 29
  AIM-INT (Month 4) | 4.33 (0.68) | 4.43 (0.56)
  AIM-INT (Month 12): number analyzed (Participants) | 52 | 29
  AIM-INT (Month 12) | 4.41 (0.57) | 4.52 (0.56)
  AIM-IMP (Baseline) | 3.97 (0.83) | 4.05 (0.76)
  AIM-IMP (Month 4): number analyzed (Participants) | 51 | 29
  AIM-IMP (Month 4) | 3.92 (0.80) | 3.86 (0.84)
  AIM-IMP (Month 12): number analyzed (Participants) | 56 | 29
  AIM-IMP (Month 12) | 4.09 (0.67) | 3.90 (1.08)

37. Secondary Outcome: Number of SSPs With Responses to ISQs Regarding Managing Delivery of APRETUDE
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, SSPs were asked about the perceived barriers to managing delivery of APRETUDE.
  Timeframe for evaluation of this outcome measure is BL, M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: At Baseline (Month 1), Month 4 and Month 12
Population: Analysis was performed on all SSPs who completed at least one survey at any timepoint. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 56 | 30
Participants
  Baseline- Management of scheduling injection appointments during correct injection windows: Extremely concerned | 3 | 2
  Baseline- Management of scheduling injection appointments during correct injection windows: Moderately concerned | 5 | 4
  Baseline- Management of scheduling injection appointments during correct injection windows: Somewhat concerned | 13 | 2
  Baseline- Management of scheduling injection appointments during correct injection windows: Slightly concerned | 5 | 7
  Baseline- Management of scheduling injection appointments during correct injection windows: Not at all concerned | 30 | 15
  Baseline- Management of rescheduling appointments during correct injection windows: Extremely concerned | 4 | 2
  Baseline- Management of rescheduling appointments during correct injection windows: Moderately concerned | 4 | 6
  Baseline- Management of rescheduling appointments during correct injection windows: Somewhat concerned | 15 | 3
  Baseline- Management of rescheduling appointments during correct injection windows: Slightly concerned | 6 | 9
  Baseline- Management of rescheduling appointments during correct injection windows: Not at all concerned | 27 | 10
  Baseline- Ability to schedule/reschedule patients who missed APRETUDE visits: Extremely concerned | 4 | 3
  Baseline- Ability to schedule/reschedule patients who missed APRETUDE visits: Moderately concerned | 5 | 4
  Baseline- Ability to schedule/reschedule patients who missed APRETUDE visits: Somewhat concerned | 16 | 5
  Baseline- Ability to schedule/reschedule patients who missed APRETUDE visits: Slightly concerned | 4 | 9
  Baseline- Ability to schedule/reschedule patients who missed APRETUDE visits: Not at all concerned | 27 | 9
  Baseline- Ability to identify and flag missed injection visits to providers (in a timely manner): Extremely concerned | 5 | 5
  Baseline- Ability to identify and flag missed injection visits to providers (in a timely manner): Moderately concerned | 5 | 5
  Baseline- Ability to identify and flag missed injection visits to providers (in a timely manner): Somewhat concerned | 15 | 4
  Baseline- Ability to identify and flag missed injection visits to providers (in a timely manner): Slightly concerned | 5 | 4
  Baseline- Ability to identify and flag missed injection visits to providers (in a timely manner): Not at all concerned | 26 | 12
  Baseline- Ability to manage patients presenting to APRETUDE appointments with other care needs: Extremely concerned | 5 | 3
  Baseline- Ability to manage patients presenting to APRETUDE appointments with other care needs: Moderately concerned | 4 | 4
  Baseline- Ability to manage patients presenting to APRETUDE appointments with other care needs: Somewhat concerned | 11 | 4
  Baseline- Ability to manage patients presenting to APRETUDE appointments with other care needs: Slightly concerned | 9 | 5
  Baseline- Ability to manage patients presenting to APRETUDE appointments with other care needs: Not at all concerned | 27 | 14
  Month 4- Management of scheduling injection appointments during correct injection windows: number analyzed (Participants) | 51 | 29
  Month 4- Management of scheduling injection appointments during correct injection windows: Extremely concerned | 2 | 2
  Month 4- Management of scheduling injection appointments during correct injection windows: Moderately concerned | 5 | 0
  Month 4- Management of scheduling injection appointments during correct injection windows: Somewhat concerned | 6 | 2
  Month 4- Management of scheduling injection appointments during correct injection windows: Slightly concerned | 3 | 4
  Month 4- Management of scheduling injection appointments during correct injection windows: Not at all concerned | 35 | 21
  Month 4- Management of rescheduling appointments during correct injection windows: number analyzed (Participants) | 51 | 29
  Month 4- Management of rescheduling appointments during correct injection windows: Extremely concerned | 2 | 2
  Month 4- Management of rescheduling appointments during correct injection windows: Moderately concerned | 5 | 1
  Month 4- Management of rescheduling appointments during correct injection windows: Somewhat concerned | 8 | 2
  Month 4- Management of rescheduling appointments during correct injection windows: Slightly concerned | 4 | 9
  Month 4- Management of rescheduling appointments during correct injection windows: Not at all concerned | 32 | 15
  Month 4- Ability to schedule/reschedule patients who missed APRETUDE visits within injection windows: number analyzed (Participants) | 51 | 29
  Month 4- Ability to schedule/reschedule patients who missed APRETUDE visits within injection windows: Extremely concerned | 1 | 2
  Month 4- Ability to schedule/reschedule patients who missed APRETUDE visits within injection windows: Moderately concerned | 5 | 1
  Month 4- Ability to schedule/reschedule patients who missed APRETUDE visits within injection windows: Somewhat concerned | 11 | 1
  Month 4- Ability to schedule/reschedule patients who missed APRETUDE visits within injection windows: Slightly concerned | 7 | 10
  Month 4- Ability to schedule/reschedule patients who missed APRETUDE visits within injection windows: Not at all concerned | 27 | 15
  Month 4- Ability to identify and flag missed injection visits to providers (in a timely manner): number analyzed (Participants) | 51 | 29
  Month 4- Ability to identify and flag missed injection visits to providers (in a timely manner): Extremely concerned | 3 | 2
  Month 4- Ability to identify and flag missed injection visits to providers (in a timely manner): Moderately concerned | 7 | 2
  Month 4- Ability to identify and flag missed injection visits to providers (in a timely manner): Somewhat concerned | 10 | 2
  Month 4- Ability to identify and flag missed injection visits to providers (in a timely manner): Slightly concerned | 6 | 7
  Month 4- Ability to identify and flag missed injection visits to providers (in a timely manner): Not at all concerned | 25 | 16
  Month 4- Ability to manage patients presenting to APRETUDE appointments with other care needs: number analyzed (Participants) | 51 | 29
  Month 4- Ability to manage patients presenting to APRETUDE appointments with other care needs: Extremely concerned | 1 | 3
  Month 4- Ability to manage patients presenting to APRETUDE appointments with other care needs: Moderately concerned | 5 | 2
  Month 4- Ability to manage patients presenting to APRETUDE appointments with other care needs: Somewhat concerned | 15 | 1
  Month 4- Ability to manage patients presenting to APRETUDE appointments with other care needs: Slightly concerned | 5 | 3
  Month 4- Ability to manage patients presenting to APRETUDE appointments with other care needs: Not at all concerned | 25 | 20
  Month 12- Management of scheduling injection appointments every 2 months during injection windows: number analyzed (Participants) | 52 | 29
  Month 12- Management of scheduling injection appointments every 2 months during injection windows: Extremely concerned | 0 | 1
  Month 12- Management of scheduling injection appointments every 2 months during injection windows: Moderately concerned | 4 | 2
  Month 12- Management of scheduling injection appointments every 2 months during injection windows: Somewhat concerned | 5 | 2
  Month 12- Management of scheduling injection appointments every 2 months during injection windows: Slightly concerned | 7 | 4
  Month 12- Management of scheduling injection appointments every 2 months during injection windows: Not at all concerned | 36 | 20
  Month 12- Management of rescheduling appointments during correct injection windows: number analyzed (Participants) | 52 | 29
  Month 12- Management of rescheduling appointments during correct injection windows: Extremely concerned | 1 | 1
  Month 12- Management of rescheduling appointments during correct injection windows: Moderately concerned | 4 | 3
  Month 12- Management of rescheduling appointments during correct injection windows: Somewhat concerned | 8 | 1
  Month 12- Management of rescheduling appointments during correct injection windows: Slightly concerned | 10 | 7
  Month 12- Management of rescheduling appointments during correct injection windows: Not at all concerned | 29 | 17
  Month 12- Ability to schedule/reschedule patients who missed APRETUDE visits: number analyzed (Participants) | 52 | 29
  Month 12- Ability to schedule/reschedule patients who missed APRETUDE visits: Extremely concerned | 2 | 1
  Month 12- Ability to schedule/reschedule patients who missed APRETUDE visits: Moderately concerned | 3 | 2
  Month 12- Ability to schedule/reschedule patients who missed APRETUDE visits: Somewhat concerned | 8 | 3
  Month 12- Ability to schedule/reschedule patients who missed APRETUDE visits: Slightly concerned | 11 | 9
  Month 12- Ability to schedule/reschedule patients who missed APRETUDE visits: Not at all concerned | 28 | 14
  Month 12- Ability to identify and flag missed injection visits to providers (in a timely manner): number analyzed (Participants) | 52 | 29
  Month 12- Ability to identify and flag missed injection visits to providers (in a timely manner): Extremely concerned | 4 | 3
  Month 12- Ability to identify and flag missed injection visits to providers (in a timely manner): Moderately concerned | 4 | 0
  Month 12- Ability to identify and flag missed injection visits to providers (in a timely manner): Somewhat concerned | 8 | 5
  Month 12- Ability to identify and flag missed injection visits to providers (in a timely manner): Slightly concerned | 10 | 9
  Month 12- Ability to identify and flag missed injection visits to providers (in a timely manner): Not at all concerned | 26 | 12
  Month 12- Ability to manage patients presenting to APRETUDE appointments with other care needs: number analyzed (Participants) | 52 | 29
  Month 12- Ability to manage patients presenting to APRETUDE appointments with other care needs: Extremely concerned | 1 | 1
  Month 12- Ability to manage patients presenting to APRETUDE appointments with other care needs: Moderately concerned | 3 | 3
  Month 12- Ability to manage patients presenting to APRETUDE appointments with other care needs: Somewhat concerned | 10 | 2
  Month 12- Ability to manage patients presenting to APRETUDE appointments with other care needs: Slightly concerned | 9 | 6
  Month 12- Ability to manage patients presenting to APRETUDE appointments with other care needs: Not at all concerned | 29 | 17

38. Secondary Outcome: Change From Baseline in AIM Score Assessed for SSPs
Description: AIM score for SSPs has 2 parts- AIM-INT that evaluates perceived intervention acceptability among SSPs and consists of 4 items (1. APRETUDE in our clinic/practice meets my approval 2. APRETUDE in our clinic/practice is appealing to me 3. I like APRETUDE in our clinic/practice 4. I welcome APRETUDE in our clinic/practice), and AIM-IMP that evaluates perceived acceptability of DI and RI approaches among SSPs and consists of 4 items (1. The implementation support has met my approval; 2. The implementation support was appealing to me; 3. I like the implementation support I have received; 4. I welcome the implementation support I have received),each with a five-point rating scale (1=completely disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, and 5=completely agree). Mean score ranges from 1 to 5 with 1=least acceptability and 5=most acceptability.
  Timeframe for evaluation is M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI) compared to BL.
Time Frame: At Month 4 and Month 12 compared to baseline (Month 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 48 | 29
Scores on a scale
  AIM-INT, Month 4 compared to BL | -0.36 (0.66) | -0.22 (0.67)
  AIM-INT, Month 12 compared to BL: number analyzed (Participants) | 40 | 26
  AIM-INT, Month 12 compared to BL | -0.33 (0.50) | -0.11 (0.74)
  AIM-IMP, Month 4 compared to BL | -0.06 (0.77) | -0.16 (0.81)
  AIM-IMP, Month 12 compared to BL: number analyzed (Participants) | 40 | 26
  AIM-IMP, Month 12 compared to BL | 0.04 (0.84) | -0.20 (1.24)

39. Secondary Outcome: Percentage of SSPs With Change From Baseline in ISQ Responses Regarding Managing Delivery of APRETUDE
Description: The ISQ used a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, SSPs were asked about the perceived barriers to managing delivery of APRETUDE (Item [I]1= Management of scheduling injection appointments during correct injection windows, I2= Management of rescheduling appointments during correct injection windows, I3= Ability to schedule/reschedule patients who missed APRETUDE visits, I4= Ability to identify and flag missed injection visits to providers (in a timely manner), I5= Ability to manage patients presenting to APRETUDE appointments with other care needs).
  Timeframe for evaluation of this outcome measure is BL, M4 and M12 (equivalent to M5 and M13 for SSPs who assessed PSPs receiving OLI). The change from baseline is calculated as a difference of percentages resulted at each timepoint as following: M4 minus (-) BL, and M12-BL.
Time Frame: At Month 4 and 12 compared to Baseline (Month 1)
Population: as for outcome 37
Measure: Number; unit: Percentage of participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 52 | 29
Percentage of participants
  Change BL to M4 - I1: Extremely concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I1: Extremely concerned | -1.4 | 0.2
  Change BL to M4 - I1: Moderately concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I1: Moderately concerned | 0.9 | -13.3
  Change BL to M4 - I1: Somewhat concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I1: Somewhat concerned | -11.4 | 0.2
  Change BL to M4 - I1: Slightly concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I1: Slightly concerned | -3.0 | -9.5
  Change BL to M4 - I1: Not at all concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I1: Not at all concerned | 15.1 | 22.4
  Change BL to M4 - I2: Extremely concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I2: Extremely concerned | -3.2 | 0.2
  Change BL to M4 - I2: Moderately concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I2: Moderately concerned | 2.7 | -16.6
  Change BL to M4 - I2: Somewhat concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I2: Somewhat concerned | -11.1 | -3.1
  Change BL to M4 - I2: Slightly concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I2: Slightly concerned | -2.9 | 1.0
  Change BL to M4 - I2: Not at all concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I2: Not at all concerned | 14.5 | 18.4
  Change BL to M4 - I3: Extremely concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I3: Extremely concerned | -5.2 | -3.1
  Change BL to M4 - I3: Moderately concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I3: Moderately concerned | 0.9 | -9.9
  Change BL to M4 - I3: Somewhat concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I3: Somewhat concerned | -7.0 | -13.2
  Change BL to M4 - I3: Slightly concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I3: Slightly concerned | 6.6 | 4.5
  Change BL to M4 - I3: Not at all concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I3: Not at all concerned | 4.7 | 21.7
  Change BL to M4 - I4: Extremely concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I4: Extremely concerned | -3.0 | -9.8
  Change BL to M4 - I4: Moderately concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I4: Moderately concerned | 4.8 | -9.8
  Change BL to M4 - I4: Somewhat concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I4: Somewhat concerned | -7.2 | -6.4
  Change BL to M4 - I4: Slightly concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I4: Slightly concerned | 2.8 | 10.8
  Change BL to M4 - I4: Not at all concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I4: Not at all concerned | 2.6 | 15.2
  Change BL to M4 - I5: Extremely concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I5: Extremely concerned | -7.0 | 0.3
  Change BL to M4 - I5: Moderately concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I5: Moderately concerned | 2.7 | -6.4
  Change BL to M4 - I5: Somewhat concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I5: Somewhat concerned | 9.8 | -9.9
  Change BL to M4 - I5: Slightly concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I5: Slightly concerned | -6.3 | -6.3
  Change BL to M4 - I5: Not at all concerned: number analyzed (Participants) | 51 | 29
  Change BL to M4 - I5: Not at all concerned | 0.8 | 22.3
  Change BL to M12 - I1: Extremely concerned | -5.4 | -3.2
  Change BL to M12 - I1: Moderately concerned | -1.2 | -6.4
  Change BL to M12 - I1: Somewhat concerned | -13.6 | 0.2
  Change BL to M12 - I1: Slightly concerned | 4.5 | -9.5
  Change BL to M12 - I1: Not at all concerned | 15.7 | 19.0
  Change BL to M12 - I2: Extremely concerned | -5.2 | -3.2
  Change BL to M12 - I2: Moderately concerned | 0.5 | -9.7
  Change BL to M12 - I2: Somewhat concerned | -11.4 | -6.6
  Change BL to M12 - I2: Slightly concerned | 8.5 | -5.9
  Change BL to M12 - I2: Not at all concerned | 7.6 | 25.3
  Change BL to M12 - I3: Extremely concerned | -3.3 | -6.6
  Change BL to M12 - I3: Moderately concerned | -3.2 | -6.4
  Change BL to M12 - I3: Somewhat concerned | -13.2 | -6.3
  Change BL to M12 - I3: Slightly concerned | 14.0 | 1.0
  Change BL to M12 - I3: Not at all concerned | 5.6 | 18.3
  Change BL to M12 - I4: Extremely concerned | -1.2 | -6.3
  Change BL to M12 - I4: Moderately concerned | -1.2 | -16.7
  Change BL to M12 - I4: Somewhat concerned | -11.4 | 3.9
  Change BL to M12 - I4: Slightly concerned | 10.3 | 17.7
  Change BL to M12 - I4: Not at all concerned | 3.6 | 1.4
  Change BL to M12 - I5: Extremely concerned | -7.0 | -6.6
  Change BL to M12 - I5: Moderately concerned | -1.4 | -3.0
  Change BL to M12 - I5: Somewhat concerned | -0.4 | -6.4
  Change BL to M12 - I5: Slightly concerned | 1.2 | 4.0
  Change BL to M12 - I5: Not at all concerned | 7.6 | 12.0

40. Secondary Outcome: Mean AIM Score Assessed for PSPs
Description: as for outcome 6
Time Frame: At Baseline (Month 1), Month 6 and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 105 | 77
Scores on a scale
  Baseline | 4.46 (0.69) | 4.41 (0.68)
  Month 6: number analyzed (Participants) | 94 | 65
  Month 6 | 4.57 (0.64) | 4.57 (0.55)
  Month 12: number analyzed (Participants) | 77 | 63
  Month 12 | 4.61 (0.63) | 4.60 (0.67)

41. Secondary Outcome: Number of PSPs With ISQ Responses Regarding Utility of Implementation Strategy at Baseline
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs were asked about the helpfulness of various knowledge materials used in learning about APRETUDE.
Time Frame: At Baseline (Month 1)
Population: Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who completed at least one ISQ survey at any timepoint. All questions were not administered to both RI and DI arms; hence only participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Very helpful | 35 | 32
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Helpful | 27 | 23
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Somewhat helpful | 12 | 10
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: A little helpful | 7 | 2
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Not at all helpful | 1 | 2
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Did not use it | 23 | 6
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Missing | 12 | 9
  Patient Brochure that helps understand the process of receiving APRETUDE injections: Very helpful | 37 | 30
  Patient Brochure that helps understand the process of receiving APRETUDE injections: Helpful | 27 | 25
  Patient Brochure that helps understand the process of receiving APRETUDE injections: Somewhat helpful | 11 | 10
  Patient Brochure that helps understand the process of receiving APRETUDE injections: A little helpful | 5 | 3
  Patient Brochure that helps understand the process of receiving APRETUDE injections: Not at all helpful | 1 | 0
  Patient Brochure that helps understand the process of receiving APRETUDE injections: Did not use it | 24 | 7
  Patient Brochure that helps understand the process of receiving APRETUDE injections: Missing | 12 | 9
  Let's talk about HIV & PrEP video that gives key facts about HIV and PrEP options (DI): number analyzed (Participants) | 117 | 0
  Let's talk about HIV & PrEP video that gives key facts about HIV and PrEP options (DI): Very helpful | 32 | 0
  Let's talk about HIV & PrEP video that gives key facts about HIV and PrEP options (DI): Helpful | 25 | 0
  Let's talk about HIV & PrEP video that gives key facts about HIV and PrEP options (DI): Somewhat helpful | 8 | 0
  Let's talk about HIV & PrEP video that gives key facts about HIV and PrEP options (DI): A little helpful | 7 | 0
  Let's talk about HIV & PrEP video that gives key facts about HIV and PrEP options (DI): Not at all helpful | 1 | 0
  Let's talk about HIV & PrEP video that gives key facts about HIV and PrEP options (DI): Did not use it | 32 | 0
  Let's talk about HIV & PrEP video that gives key facts about HIV and PrEP options (DI): Missing | 12 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): number analyzed (Participants) | 117 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Very helpful | 30 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Helpful | 22 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Somewhat helpful | 8 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): A little helpful | 6 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Not at all helpful | 1 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Did not use it | 38 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Missing | 12 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): number analyzed (Participants) | 117 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Very helpful | 30 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Helpful | 25 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Somewhat helpful | 7 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): A little helpful | 5 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Not at all helpful | 0 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Did not use it | 38 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Missing | 12 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): number analyzed (Participants) | 117 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Very helpful | 26 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Helpful | 23 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Somewhat helpful | 9 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): A little helpful | 6 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Not at all helpful | 0 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Did not use it | 41 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Missing | 12 | 0
  The study website to access APRETDUE information (RI): number analyzed (Participants) | 0 | 84
  The study website to access APRETDUE information (RI): Very helpful | 0 | 28
  The study website to access APRETDUE information (RI): Helpful | 0 | 19
  The study website to access APRETDUE information (RI): Somewhat helpful | 0 | 13
  The study website to access APRETDUE information (RI): A little helpful | 0 | 4
  The study website to access APRETDUE information (RI): Not at all helpful | 0 | 0
  The study website to access APRETDUE information (RI): Did not use it | 0 | 11
  The study website to access APRETDUE information (RI): Missing | 0 | 9
  The study app to access APRETUDE information (DI): number analyzed (Participants) | 117 | 0
  The study app to access APRETUDE information (DI): Very helpful | 23 | 0
  The study app to access APRETUDE information (DI): Helpful | 22 | 0
  The study app to access APRETUDE information (DI): Somewhat helpful | 12 | 0
  The study app to access APRETUDE information (DI): A little helpful | 6 | 0
  The study app to access APRETUDE information (DI): Not at all helpful | 0 | 0
  The study app to access APRETUDE information (DI): Did not use it | 42 | 0
  The study app to access APRETUDE information (DI): Missing | 12 | 0

42. Secondary Outcome: Number of PSPs With ISQ Responses Regarding Utility of Implementation Strategy at Month 6
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs were asked about the helpfulness of various knowledge materials used in learning about APRETUDE.
  Timeframe for evaluation of this outcome measure is M6 (equivalent to M7 for PSPs who received OLI).
Time Frame: At Month 6
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Very helpful | 28 | 24
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Helpful | 17 | 17
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Somewhat helpful | 18 | 6
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: A little helpful | 3 | 0
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Not at all helpful | 1 | 0
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Did not receive/Did not use it | 25 | 16
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Missing | 25 | 21
  Patient Brochure helps understand the process of receiving APRETUDE injections: Very helpful | 29 | 21
  Patient Brochure helps understand the process of receiving APRETUDE injections: Helpful | 17 | 18
  Patient Brochure helps understand the process of receiving APRETUDE injections: Somewhat helpful | 14 | 7
  Patient Brochure helps understand the process of receiving APRETUDE injections: A little helpful | 2 | 1
  Patient Brochure helps understand the process of receiving APRETUDE injections: Not at all helpful | 1 | 0
  Patient Brochure helps understand the process of receiving APRETUDE injections: Did not receive/Did not use it | 29 | 16
  Patient Brochure helps understand the process of receiving APRETUDE injections: Missing | 25 | 21
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): number analyzed (Participants) | 117 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Very helpful | 27 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Helpful | 19 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Somewhat helpful | 8 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): A little helpful | 5 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Not at all helpful | 1 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Did not receive/Did not use it | 32 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Missing | 25 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): number analyzed (Participants) | 117 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Very helpful | 23 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Helpful | 20 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Somewhat helpful | 8 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): A little helpful | 5 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Not at all helpful | 2 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Did not receive/Did not use it | 34 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Missing | 25 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): number analyzed (Participants) | 117 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Very helpful | 26 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Helpful | 16 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Somewhat helpful | 9 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): A little helpful | 4 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Not at all helpful | 1 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Did not receive/Did not use it | 36 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Missing | 25 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): number analyzed (Participants) | 117 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Very helpful | 22 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Helpful | 15 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Somewhat helpful | 10 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): A little helpful | 6 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Not at all helpful | 1 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Did not receive/Did not use it | 38 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Missing | 25 | 0
  The study website to access APRETDUE information (RI): number analyzed (Participants) | 0 | 84
  The study website to access APRETDUE information (RI): Very helpful | 0 | 21
  The study website to access APRETDUE information (RI): Helpful | 0 | 16
  The study website to access APRETDUE information (RI): Somewhat helpful | 0 | 8
  The study website to access APRETDUE information (RI): A little helpful | 0 | 2
  The study website to access APRETDUE information (RI): Not at all helpful | 0 | 1
  The study website to access APRETDUE information (RI): Did not receive/Did not use it | 0 | 15
  The study website to access APRETDUE information (RI): Missing | 0 | 21
  The study app to access APRETUDE information (DI): number analyzed (Participants) | 117 | 0
  The study app to access APRETUDE information (DI): Very helpful | 24 | 0
  The study app to access APRETUDE information (DI): Helpful | 17 | 0
  The study app to access APRETUDE information (DI): Somewhat helpful | 15 | 0
  The study app to access APRETUDE information (DI): A little helpful | 8 | 0
  The study app to access APRETUDE information (DI): Not at all helpful | 5 | 0
  The study app to access APRETUDE information (DI): Did not receive/Did not use it | 23 | 0
  The study app to access APRETUDE information (DI): Missing | 25 | 0
  Important safety information document details safety information relating to APRETUDE: Very helpful | 26 | 19
  Important safety information document details safety information relating to APRETUDE: Helpful | 17 | 18
  Important safety information document details safety information relating to APRETUDE: Somewhat helpful | 11 | 9
  Important safety information document details safety information relating to APRETUDE: A little helpful | 8 | 0
  Important safety information document details safety information relating to APRETUDE: Not at all helpful | 2 | 1
  Important safety information document details safety information relating to APRETUDE: Did not receive/Did not use it | 28 | 16
  Important safety information document details safety information relating to APRETUDE: Missing | 25 | 21
  Important facts document details important facts relating to APRETUDE: Very helpful | 26 | 19
  Important facts document details important facts relating to APRETUDE: Helpful | 19 | 17
  Important facts document details important facts relating to APRETUDE: Somewhat helpful | 10 | 9
  Important facts document details important facts relating to APRETUDE: A little helpful | 4 | 1
  Important facts document details important facts relating to APRETUDE: Not at all helpful | 1 | 1
  Important facts document details important facts relating to APRETUDE: Did not receive/Did not use it | 32 | 16
  Important facts document details important facts relating to APRETUDE: Missing | 25 | 21
  A flyer on PrEP options (DI): number analyzed (Participants) | 117 | 0
  A flyer on PrEP options (DI): Very helpful | 22 | 0
  A flyer on PrEP options (DI): Helpful | 16 | 0
  A flyer on PrEP options (DI): Somewhat helpful | 9 | 0
  A flyer on PrEP options (DI): A little helpful | 2 | 0
  A flyer on PrEP options (DI): Not at all helpful | 2 | 0
  A flyer on PrEP options (DI): Did not receive/Did not use it | 41 | 0
  A flyer on PrEP options (DI): Missing | 25 | 0

43. Secondary Outcome: Number of PSPs With ISQ Responses Regarding Utility of Implementation Strategy at Month 12
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs were asked about the helpfulness of various knowledge materials used in learning about APRETUDE.
  Timeframe for evaluation of this outcome measure is M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: At Month 12
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Very helpful | 23 | 24
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Helpful | 26 | 14
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Somewhat helpful | 5 | 8
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: A little helpful | 5 | 2
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Not at all helpful | 0 | 2
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Did not receive/Did not use it | 18 | 13
  Getting Started Brochure that gives an overview of how to get started with APRETUDE: Missing | 40 | 21
  Patient Brochure helps understand the process of receiving APRETUDE injections: Very helpful | 22 | 22
  Patient Brochure helps understand the process of receiving APRETUDE injections: Helpful | 27 | 14
  Patient Brochure helps understand the process of receiving APRETUDE injections: Somewhat helpful | 6 | 10
  Patient Brochure helps understand the process of receiving APRETUDE injections: A little helpful | 4 | 3
  Patient Brochure helps understand the process of receiving APRETUDE injections: Not at all helpful | 0 | 1
  Patient Brochure helps understand the process of receiving APRETUDE injections: Did not receive/Did not use it | 18 | 13
  Patient Brochure helps understand the process of receiving APRETUDE injections: Missing | 40 | 21
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): number analyzed (Participants) | 117 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Very helpful | 25 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Helpful | 20 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Somewhat helpful | 6 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): A little helpful | 5 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Not at all helpful | 0 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Did not receive/Did not use it | 21 | 0
  Let's talk about HIV & PrEP video gives key facts about HIV and PrEP options (DI): Missing | 40 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): number analyzed (Participants) | 117 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Very helpful | 25 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Helpful | 18 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Somewhat helpful | 7 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): A little helpful | 3 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Not at all helpful | 0 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Did not receive/Did not use it | 24 | 0
  The APRETUDE Myths and Facts video, the game show video addressing common myths about APRETUDE (DI): Missing | 40 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): number analyzed (Participants) | 117 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Very helpful | 26 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Helpful | 17 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Somewhat helpful | 6 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): A little helpful | 5 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Not at all helpful | 0 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Did not receive/Did not use it | 23 | 0
  The What to Expect video which shows what to expect during the APRETUDE process (DI): Missing | 40 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): number analyzed (Participants) | 117 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Very helpful | 22 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Helpful | 20 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Somewhat helpful | 8 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): A little helpful | 3 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Not at all helpful | 0 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Did not receive/Did not use it | 24 | 0
  The ViiV Connect Video tells about the ViiV Connect program and frequently asked questions (DI): Missing | 40 | 0
  The study website to access APRETDUE information (RI): number analyzed (Participants) | 0 | 84
  The study website to access APRETDUE information (RI): Very helpful | 0 | 19
  The study website to access APRETDUE information (RI): Helpful | 0 | 16
  The study website to access APRETDUE information (RI): Somewhat helpful | 0 | 7
  The study website to access APRETDUE information (RI): A little helpful | 0 | 7
  The study website to access APRETDUE information (RI): Not at all helpful | 0 | 1
  The study website to access APRETDUE information (RI): Did not receive/Did not use it | 0 | 13
  The study website to access APRETDUE information (RI): Missing | 0 | 21
  The study app/website to access APRETUDE information - the Pillar Spot (DI): number analyzed (Participants) | 117 | 0
  The study app/website to access APRETUDE information - the Pillar Spot (DI): Very helpful | 22 | 0
  The study app/website to access APRETUDE information - the Pillar Spot (DI): Helpful | 19 | 0
  The study app/website to access APRETUDE information - the Pillar Spot (DI): Somewhat helpful | 9 | 0
  The study app/website to access APRETUDE information - the Pillar Spot (DI): A little helpful | 8 | 0
  The study app/website to access APRETUDE information - the Pillar Spot (DI): Not at all helpful | 1 | 0
  The study app/website to access APRETUDE information - the Pillar Spot (DI): Did not receive/Did not use it | 18 | 0
  The study app/website to access APRETUDE information - the Pillar Spot (DI): Missing | 40 | 0
  Important safety information document details safety information relating to APRETUDE: Very helpful | 22 | 19
  Important safety information document details safety information relating to APRETUDE: Helpful | 22 | 17
  Important safety information document details safety information relating to APRETUDE: Somewhat helpful | 9 | 9
  Important safety information document details safety information relating to APRETUDE: A little helpful | 2 | 5
  Important safety information document details safety information relating to APRETUDE: Not at all helpful | 0 | 1
  Important safety information document details safety information relating to APRETUDE: Did not receive/Did not use it | 22 | 12
  Important safety information document details safety information relating to APRETUDE: Missing | 40 | 21
  Important facts document details important facts relating to APRETUDE: Very helpful | 21 | 20
  Important facts document details important facts relating to APRETUDE: Helpful | 23 | 16
  Important facts document details important facts relating to APRETUDE: Somewhat helpful | 8 | 7
  Important facts document details important facts relating to APRETUDE: A little helpful | 1 | 6
  Important facts document details important facts relating to APRETUDE: Not at all helpful | 0 | 1
  Important facts document details important facts relating to APRETUDE: Did not receive/Did not use it | 24 | 13
  Important facts document details important facts relating to APRETUDE: Missing | 40 | 21
  A flyer on PrEP options: Very helpful | 22 | 19
  A flyer on PrEP options: Helpful | 17 | 14
  A flyer on PrEP options: Somewhat helpful | 8 | 7
  A flyer on PrEP options: A little helpful | 2 | 5
  A flyer on PrEP options: Not at all helpful | 1 | 1
  A flyer on PrEP options: Did not receive/Did not use it | 27 | 17
  A flyer on PrEP options: Missing | 40 | 21

44. Secondary Outcome: Change From Baseline in Mean AIM Score in PSPs
Description: as for outcome 12
Time Frame: At Month 6 and Month 12 compared to baseline (Month 1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Scores on a scale
  Month 6 compared to BL: number analyzed (Participants) | 87 | 61
  Month 6 compared to BL | 0.17 (0.66) | 0.20 (0.72)
  Month 12 compared to BL: number analyzed (Participants) | 71 | 59
  Month 12 compared to BL | 0.27 (0.63) | 0.19 (0.87)

45. Secondary Outcome: Percentage of PSPs With Change From Baseline in ISQ Responses Under Implementation Strategy
Description: In this outcome measure, usong the ISQ, PSPs were asked about the helpfulness of various knowledge materials (I1= Getting Started Brochure that gives an overview of how to get started with APRETUDE, I2 = Patient Brochure helps understand the process of receiving APRETUDE, I3 = HIV & PrEP video gives key facts about HIV and PrEP options (DI), I4 = APRETUDE Myths and Facts video, addressing common myths about APRETUDE (DI), I5 = The What to Expect video which shows what to expect during the APRETUDE process (DI), I6 = The ViiV Connect program Video and frequently asked questions (DI), I7 = The study website to access APRETDUE information (RI), I8 = The study app to access APRETUDE information (DI). Timeframe for evaluation of this outcome measure is M6 and M12 (equivalent to M7 and M13 for PSPs who received OLI). The change from baseline is calculated as a difference of percentages resulted at each timepoint as following: M6 minus (-) BL, and M12-BL.
Time Frame: At Month 6 and Month 12 compared to Baseline (Month 1)
Population: Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who completed at least one ISQ survey at any timepoint. All questions were not administered to both RI and DI arms; hence, certain Rows have 0 participants analyzed within each Arm/Group.
Measure: Number; unit: Percentage of participants
Groups:
- DI - PSP: Men who have sex with men (MSM) and transgender men (TGM) who were HIV negative as PSPs received APRETUDE injection (Direct to Injection - DTI) and had the choice to receive an optional cabotegravir tablets as oral lead in (OLI). PSPs had access to enhanced toolkits and digital health implementation supports.
- RI - PSP: MSM and transgender men who were HIV negative as PSPs received APRETUDE injection (DTI) and had the choice to use an optional cabotegravir tablets as OLI. PSPs had access to standard toolkits for APRETUDE to use as needed.
Arm/Group | DI - PSP | RI - PSP
Number analyzed (Participants) | 92 | 63
Percentage of participants
  Change BL to M6 - I1: Very helpful | -2.9 | -4.6
  Change BL to M6 - I1: Helpful | -7.2 | -3.7
  Change BL to M6 - I1: Somewhat helpful | 8.1 | -3.8
  Change BL to M6 - I1: A little helpful | -3.4 | -2.7
  Change BL to M6 - I1: Not at all helpful | 0.1 | -2.7
  Change BL to M6 - I1: I did not use it | 5.3 | 17.4
  Change BL to M6 - I2: Very helpful | -3.7 | -6.7
  Change BL to M6 - I2: Helpful | -7.2 | -4.8
  Change BL to M6 - I2: Somewhat helpful | 4.7 | -2.2
  Change BL to M6 - I2: A little helpful | -2.6 | -2.4
  Change BL to M6 - I2: Not at all helpful | 0.1 | 0.0
  Change BL to M6 - I2: I did not use it | 8.7 | 16.1
  Change BL to M6 - I3: Very helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I3: Very helpful | -1.1 |
  Change BL to M6 - I3: Helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I3: Helpful | -3.2 |
  Change BL to M6 - I3: Somewhat helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I3: Somewhat helpful | 1.1 |
  Change BL to M6 - I3: A little helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I3: A little helpful | -1.2 |
  Change BL to M6 - I3: Not at all helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I3: Not at all helpful | 0.1 |
  Change BL to M6 - I3: I did not use it: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I3: I did not use it | 4.3 |
  Change BL to M6 - I4: Very helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I4: Very helpful | -3.6 |
  Change BL to M6 - I4: Helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I4: Helpful | 0.8 |
  Change BL to M6 - I4: Somewhat helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I4: Somewhat helpful | 1.1 |
  Change BL to M6 - I4: A little helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I4: A little helpful | -0.3 |
  Change BL to M6 - I4: Not at all helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I4: Not at all helpful | 1.2 |
  Change BL to M6 - I4: I did not use it: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I4: I did not use it | 0.8 |
  Change BL to M6 - I5: Very helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I5: Very helpful | -0.3 |
  Change BL to M6 - I5: Helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I5: Helpful | -6.4 |
  Change BL to M6 - I5: Somewhat helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I5: Somewhat helpful | 3.1 |
  Change BL to M6 - I5: A little helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I5: A little helpful | -0.4 |
  Change BL to M6 - I5: Not at all helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I5: Not at all helpful | 1.1 |
  Change BL to M6 - I5: I did not use it: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I5: I did not use it | 2.9 |
  Change BL to M6 - I6: Very helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I6: Very helpful | -0.8 |
  Change BL to M6 - I6: Helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I6: Helpful | -5.6 |
  Change BL to M6 - I6: Somewhat helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I6: Somewhat helpful | 2.3 |
  Change BL to M6 - I6: A little helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I6: A little helpful | 0.8 |
  Change BL to M6 - I6: Not at all helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I6: Not at all helpful | 1.1 |
  Change BL to M6 - I6: I did not use it: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I6: I did not use it | 2.3 |
  Change BL to M6 - I7: Very helpful: number analyzed (Participants) | 0 | 63
  Change BL to M6 - I7: Very helpful |  | -4.0
  Change BL to M6 - I7: Helpful: number analyzed (Participants) | 0 | 63
  Change BL to M6 - I7: Helpful |  | 0.1
  Change BL to M6 - I7: Somewhat helpful: number analyzed (Participants) | 0 | 63
  Change BL to M6 - I7: Somewhat helpful |  | -4.6
  Change BL to M6 - I7: A little helpful: number analyzed (Participants) | 0 | 63
  Change BL to M6 - I7: A little helpful |  | -2.2
  Change BL to M6 - I7: Not at all helpful: number analyzed (Participants) | 0 | 63
  Change BL to M6 - I7: Not at all helpful |  | 1.6
  Change BL to M6 - I7: I did not use it: number analyzed (Participants) | 0 | 63
  Change BL to M6 - I7: I did not use it |  | 9.1
  Change BL to M6 - I8: Very helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I8: Very helpful | 4.2 |
  Change BL to M6 - I8: Helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I8: Helpful | -2.5 |
  Change BL to M6 - I8: Somewhat helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I8: Somewhat helpful | 4.9 |
  Change BL to M6 - I8: A little helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I8: A little helpful | 3.0 |
  Change BL to M6 - I8: Not at all helpful: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I8: Not at all helpful | 5.4 |
  Change BL to M6 - I8: I did not use it: number analyzed (Participants) | 92 | 0
  Change BL to M6 - I8: I did not use it | -15.0 |
  Change BL to M12 - I1: Very helpful: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I1: Very helpful | -3.5 | -4.6
  Change BL to M12 - I1: Helpful: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I1: Helpful | 8.1 | -8.4
  Change BL to M12 - I1: Somewhat helpful: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I1: Somewhat helpful | -4.9 | -0.6
  Change BL to M12 - I1: A little helpful: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I1: A little helpful | -0.2 | 0.5
  Change BL to M12 - I1: Not at all helpful: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I1: Not at all helpful | -1.0 | 0.5
  Change BL to M12 - I1: I did not use it: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I1: I did not use it | 1.5 | 12.6
  Change BL to M12 - I2: Very helpful: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I2: Very helpful | -6.7 | -5.1
  Change BL to M12 - I2: Helpful: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I2: Helpful | 9.4 | -11.1
  Change BL to M12 - I2: Somewhat helpful: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I2: Somewhat helpful | -2.7 | 2.5
  Change BL to M12 - I2: A little helpful: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I2: A little helpful | 0.4 | 0.8
  Change BL to M12 - I2: Not at all helpful: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I2: Not at all helpful | -1.0 | 1.6
  Change BL to M12 - I2: I did not use it: number analyzed (Participants) | 77 | 63
  Change BL to M12 - I2: I did not use it | 0.5 | 11.3
  Change BL to M12 - I3: Very helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I3: Very helpful | 2.0 |
  Change BL to M12 - I3: Helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I3: Helpful | 2.2 |
  Change BL to M12 - I3: Somewhat helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I3: Somewhat helpful | 0.2 |
  Change BL to M12 - I3: A little helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I3: A little helpful | -0.2 |
  Change BL to M12 - I3: Not at all helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I3: Not at all helpful | -1.0 |
  Change BL to M12 - I3: I did not use it: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I3: I did not use it | -3.2 |
  Change BL to M12 - I4: Very helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I4: Very helpful | 3.9 |
  Change BL to M12 - I4: Helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I4: Helpful | 2.4 |
  Change BL to M12 - I4: Somewhat helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I4: Somewhat helpful | 1.5 |
  Change BL to M12 - I4: A little helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I4: A little helpful | -1.8 |
  Change BL to M12 - I4: Not at all helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I4: Not at all helpful | -1.0 |
  Change BL to M12 - I4: I did not use it: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I4: I did not use it | -5.0 |
  Change BL to M12 - I5: Very helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I5: Very helpful | 5.2 |
  Change BL to M12 - I5: Helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I5: Helpful | -1.7 |
  Change BL to M12 - I5: Somewhat helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I5: Somewhat helpful | 1.1 |
  Change BL to M12 - I5: A little helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I5: A little helpful | 1.7 |
  Change BL to M12 - I5: Not at all helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I5: Not at all helpful | 0.0 |
  Change BL to M12 - I5: I did not use it: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I5: I did not use it | -6.3 |
  Change BL to M12 - I6: Very helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I6: Very helpful | 3.8 |
  Change BL to M12 - I6: Helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I6: Helpful | 4.1 |
  Change BL to M12 - I6: Somewhat helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I6: Somewhat helpful | 1.8 |
  Change BL to M12 - I6: A little helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I6: A little helpful | -1.8 |
  Change BL to M12 - I6: Not at all helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I6: Not at all helpful | 0.0 |
  Change BL to M12 - I6: I did not use it: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I6: I did not use it | -7.9 |
  Change BL to M12 - I7: Very helpful: number analyzed (Participants) | 0 | 63
  Change BL to M12 - I7: Very helpful |  | -7.2
  Change BL to M12 - I7: Helpful: number analyzed (Participants) | 0 | 63
  Change BL to M12 - I7: Helpful |  | 0.1
  Change BL to M12 - I7: Somewhat helpful: number analyzed (Participants) | 0 | 63
  Change BL to M12 - I7: Somewhat helpful |  | -6.2
  Change BL to M12 - I7: A little helpful: number analyzed (Participants) | 0 | 63
  Change BL to M12 - I7: A little helpful |  | 5.8
  Change BL to M12 - I7: Not at all helpful: number analyzed (Participants) | 0 | 63
  Change BL to M12 - I7: Not at all helpful |  | 1.6
  Change BL to M12 - I7: I did not use it: number analyzed (Participants) | 0 | 24
  Change BL to M12 - I7: I did not use it |  | 6.0
  Change BL to M12 - I8: Very helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I8: Very helpful | 6.7 |
  Change BL to M12 - I8: Helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I8: Helpful | 3.7 |
  Change BL to M12 - I8: Somewhat helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I8: Somewhat helpful | 0.3 |
  Change BL to M12 - I8: A little helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I8: A little helpful | 4.7 |
  Change BL to M12 - I8: Not at all helpful: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I8: Not at all helpful | 1.3 |
  Change BL to M12 - I8: I did not use it: number analyzed (Participants) | 77 | 0
  Change BL to M12 - I8: I did not use it | -16.6 |

46. Secondary Outcome: Number of SSPs That Respond in Agreement on Relevant Items on the ISQ That Each Implementation Strategy is Fit for Use
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, SSPs were asked about the usefulness of various implementation strategies used for implementing APRETUDE in their clinic/practice.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on SSPs who completed at least one survey at any timepoint. All questions were not administered to both RI and DI arms; hence only participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 52 | 29
Participants
  Frequently Asked Questions Brochure: number analyzed (Participants) | 19 | 12
  Frequently Asked Questions Brochure: Not at all useful | 1 | 0
  Frequently Asked Questions Brochure: A little useful | 3 | 1
  Frequently Asked Questions Brochure: Somewhat useful | 5 | 1
  Frequently Asked Questions Brochure: Useful | 5 | 8
  Frequently Asked Questions Brochure: Very Useful | 5 | 2
  Readiness Consideration: number analyzed (Participants) | 16 | 11
  Readiness Consideration: Not at all useful | 0 | 0
  Readiness Consideration: A little useful | 2 | 0
  Readiness Consideration: Somewhat useful | 3 | 2
  Readiness Consideration: Useful | 5 | 7
  Readiness Consideration: Very Useful | 6 | 2
  Get Started Overview-Init/Adm Guide: number analyzed (Participants) | 19 | 11
  Get Started Overview-Init/Adm Guide: Not at all useful | 0 | 0
  Get Started Overview-Init/Adm Guide: A little useful | 3 | 0
  Get Started Overview-Init/Adm Guide: Somewhat useful | 4 | 2
  Get Started Overview-Init/Adm Guide: Useful | 6 | 7
  Get Started Overview-Init/Adm Guide: Very Useful | 6 | 2
  Injection Education Video: number analyzed (Participants) | 28 | 18
  Injection Education Video: Not at all useful | 0 | 0
  Injection Education Video: A little useful | 0 | 0
  Injection Education Video: Somewhat useful | 5 | 5
  Injection Education Video: Useful | 8 | 7
  Injection Education Video: Very Useful | 15 | 6
  Provider Website- location where all materials and videos on APRETUDE are located (RI): number analyzed (Participants) | 0 | 13
  Provider Website- location where all materials and videos on APRETUDE are located (RI): Not at all useful | 0 | 2
  Provider Website- location where all materials and videos on APRETUDE are located (RI): A little useful | 0 | 0
  Provider Website- location where all materials and videos on APRETUDE are located (RI): Somewhat useful | 0 | 2
  Provider Website- location where all materials and videos on APRETUDE are located (RI): Useful | 0 | 8
  Provider Website- location where all materials and videos on APRETUDE are located (RI): Very Useful | 0 | 1
  Patient Materials: number analyzed (Participants) | 21 | 15
  Patient Materials: Not at all useful | 0 | 0
  Patient Materials: A little useful | 3 | 0
  Patient Materials: Somewhat useful | 3 | 2
  Patient Materials: Useful | 7 | 10
  Patient Materials: Very Useful | 8 | 3
  Implementation Guidance Video (DI): number analyzed (Participants) | 17 | 0
  Implementation Guidance Video (DI): Not at all useful | 0 | 0
  Implementation Guidance Video (DI): A little useful | 2 | 0
  Implementation Guidance Video (DI): Somewhat useful | 2 | 0
  Implementation Guidance Video (DI): Useful | 9 | 0
  Implementation Guidance Video (DI): Very Useful | 4 | 0
  Appointment Scheduler: number analyzed (Participants) | 15 | 7
  Appointment Scheduler: Not at all useful | 1 | 0
  Appointment Scheduler: A little useful | 0 | 0
  Appointment Scheduler: Somewhat useful | 2 | 0
  Appointment Scheduler: Useful | 6 | 5
  Appointment Scheduler: Very Useful | 6 | 2
  Pre-scheduled Appointment Guidance (DI): number analyzed (Participants) | 15 | 0
  Pre-scheduled Appointment Guidance (DI): Not at all useful | 0 | 0
  Pre-scheduled Appointment Guidance (DI): A little useful | 0 | 0
  Pre-scheduled Appointment Guidance (DI): Somewhat useful | 3 | 0
  Pre-scheduled Appointment Guidance (DI): Useful | 6 | 0
  Pre-scheduled Appointment Guidance (DI): Very Useful | 6 | 0
  Designated Injection Days Guidance (DI): number analyzed (Participants) | 15 | 0
  Designated Injection Days Guidance (DI): Not at all useful | 0 | 0
  Designated Injection Days Guidance (DI): A little useful | 1 | 0
  Designated Injection Days Guidance (DI): Somewhat useful | 5 | 0
  Designated Injection Days Guidance (DI): Useful | 7 | 0
  Designated Injection Days Guidance (DI): Very Useful | 2 | 0
  Drop-in Injection Visits Guidance (DI): number analyzed (Participants) | 12 | 0
  Drop-in Injection Visits Guidance (DI): Not at all useful | 0 | 0
  Drop-in Injection Visits Guidance (DI): A little useful | 0 | 0
  Drop-in Injection Visits Guidance (DI): Somewhat useful | 4 | 0
  Drop-in Injection Visits Guidance (DI): Useful | 4 | 0
  Drop-in Injection Visits Guidance (DI): Very Useful | 4 | 0
  Transport Support to Patient Appt (DI): number analyzed (Participants) | 20 | 0
  Transport Support to Patient Appt (DI): Not at all useful | 0 | 0
  Transport Support to Patient Appt (DI): A little useful | 0 | 0
  Transport Support to Patient Appt (DI): Somewhat useful | 4 | 0
  Transport Support to Patient Appt (DI): Useful | 5 | 0
  Transport Support to Patient Appt (DI): Very Useful | 11 | 0
  Monthly Implement Facilitation Call (DI): number analyzed (Participants) | 24 | 0
  Monthly Implement Facilitation Call (DI): Not at all useful | 2 | 0
  Monthly Implement Facilitation Call (DI): A little useful | 0 | 0
  Monthly Implement Facilitation Call (DI): Somewhat useful | 5 | 0
  Monthly Implement Facilitation Call (DI): Useful | 9 | 0
  Monthly Implement Facilitation Call (DI): Very Useful | 8 | 0
  Group Implement Facilitation Calls (DI): number analyzed (Participants) | 24 | 0
  Group Implement Facilitation Calls (DI): Not at all useful | 1 | 0
  Group Implement Facilitation Calls (DI): A little useful | 1 | 0
  Group Implement Facilitation Calls (DI): Somewhat useful | 5 | 0
  Group Implement Facilitation Calls (DI): Useful | 8 | 0
  Group Implement Facilitation Calls (DI): Very Useful | 9 | 0
  Document on How Discuss Sex Health (DI): number analyzed (Participants) | 14 | 0
  Document on How Discuss Sex Health (DI): Not at all useful | 0 | 0
  Document on How Discuss Sex Health (DI): A little useful | 1 | 0
  Document on How Discuss Sex Health (DI): Somewhat useful | 3 | 0
  Document on How Discuss Sex Health (DI): Useful | 6 | 0
  Document on How Discuss Sex Health (DI): Very Useful | 4 | 0
  PILLAR Spot (DI): number analyzed (Participants) | 34 | 0
  PILLAR Spot (DI): Not at all useful | 1 | 0
  PILLAR Spot (DI): A little useful | 3 | 0
  PILLAR Spot (DI): Somewhat useful | 7 | 0
  PILLAR Spot (DI): Useful | 13 | 0
  PILLAR Spot (DI): Very Useful | 10 | 0

47. Secondary Outcome: Number of PSPs That Respond in Agreement on Relevant Items on the ISQ That Each Implementation Strategy is Fit for Use
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs were asked about how useful various implementation strategies have been in supporting them while taking APRETUDE.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  Brochures and other print materials to educate you on APRETUDE: number analyzed (Participants) | 49 | 35
  Brochures and other print materials to educate you on APRETUDE: Not at all useful | 1 | 0
  Brochures and other print materials to educate you on APRETUDE: Not very useful | 2 | 1
  Brochures and other print materials to educate you on APRETUDE: Somewhat useful | 10 | 10
  Brochures and other print materials to educate you on APRETUDE: Useful | 23 | 12
  Brochures and other print materials to educate you on APRETUDE: Extremely useful | 13 | 12
  Videos to educate you on HIV, PrEP, APRETUDE materials (DI): number analyzed (Participants) | 40 | 0
  Videos to educate you on HIV, PrEP, APRETUDE materials (DI): Not at all useful | 1 | 0
  Videos to educate you on HIV, PrEP, APRETUDE materials (DI): Not very useful | 1 | 0
  Videos to educate you on HIV, PrEP, APRETUDE materials (DI): Somewhat useful | 8 | 0
  Videos to educate you on HIV, PrEP, APRETUDE materials (DI): Useful | 21 | 0
  Videos to educate you on HIV, PrEP, APRETUDE materials (DI): Extremely useful | 9 | 0
  A digital calendar specifically made for APRETUDE to help plan injections, found on Pillar Spot (DI): number analyzed (Participants) | 15 | 0
  A digital calendar specifically made for APRETUDE to help plan injections, found on Pillar Spot (DI): Not at all useful | 2 | 0
  A digital calendar specifically made for APRETUDE to help plan injections, found on Pillar Spot (DI): Not very useful | 0 | 0
  A digital calendar specifically made for APRETUDE to help plan injections, found on Pillar Spot (DI): Somewhat useful | 3 | 0
  A digital calendar specifically made for APRETUDE to help plan injections, found on Pillar Spot (DI): Useful | 6 | 0
  A digital calendar specifically made for APRETUDE to help plan injections, found on Pillar Spot (DI): Extremely useful | 4 | 0
  Reminders about injections: number analyzed (Participants) | 65 | 51
  Reminders about injections: Not at all useful | 3 | 0
  Reminders about injections: Not very useful | 2 | 0
  Reminders about injections: Somewhat useful | 5 | 3
  Reminders about injections: Useful | 25 | 22
  Reminders about injections: Extremely useful | 30 | 26
  Having video or telephone appointments with your doctor: number analyzed (Participants) | 17 | 16
  Having video or telephone appointments with your doctor: Not at all useful | 1 | 0
  Having video or telephone appointments with your doctor: Not very useful | 0 | 0
  Having video or telephone appointments with your doctor: Somewhat useful | 3 | 1
  Having video or telephone appointments with your doctor: Useful | 7 | 7
  Having video or telephone appointments with your doctor: Extremely useful | 6 | 8
  Sending chats or texts to your doctor on the Pillar Spot (DI): number analyzed (Participants) | 23 | 0
  Sending chats or texts to your doctor on the Pillar Spot (DI): Not at all useful | 1 | 0
  Sending chats or texts to your doctor on the Pillar Spot (DI): Not very useful | 0 | 0
  Sending chats or texts to your doctor on the Pillar Spot (DI): Somewhat useful | 3 | 0
  Sending chats or texts to your doctor on the Pillar Spot (DI): Useful | 11 | 0
  Sending chats or texts to your doctor on the Pillar Spot (DI): Extremely useful | 8 | 0
  Having a nurse come home to conduct your HIV test (DI): number analyzed (Participants) | 5 | 0
  Having a nurse come home to conduct your HIV test (DI): Not at all useful | 1 | 0
  Having a nurse come home to conduct your HIV test (DI): Not very useful | 0 | 0
  Having a nurse come home to conduct your HIV test (DI): Somewhat useful | 1 | 0
  Having a nurse come home to conduct your HIV test (DI): Useful | 2 | 0
  Having a nurse come home to conduct your HIV test (DI): Extremely useful | 1 | 0
  Having a nurse come home to give your injection (DI): number analyzed (Participants) | 5 | 0
  Having a nurse come home to give your injection (DI): Not at all useful | 1 | 0
  Having a nurse come home to give your injection (DI): Not very useful | 0 | 0
  Having a nurse come home to give your injection (DI): Somewhat useful | 1 | 0
  Having a nurse come home to give your injection (DI): Useful | 2 | 0
  Having a nurse come home to give your injection (DI): Extremely useful | 1 | 0
  Receiving transportation to the clinic/doctor's office for your injection (DI): number analyzed (Participants) | 22 | 0
  Receiving transportation to the clinic/doctor's office for your injection (DI): Not at all useful | 1 | 0
  Receiving transportation to the clinic/doctor's office for your injection (DI): Not very useful | 0 | 0
  Receiving transportation to the clinic/doctor's office for your injection (DI): Somewhat useful | 2 | 0
  Receiving transportation to the clinic/doctor's office for your injection (DI): Useful | 4 | 0
  Receiving transportation to the clinic/doctor's office for your injection (DI): Extremely useful | 15 | 0
  A website/app to access APRETUDE information- the Pillar Spot (DI): number analyzed (Participants) | 32 | 0
  A website/app to access APRETUDE information- the Pillar Spot (DI): Not at all useful | 2 | 0
  A website/app to access APRETUDE information- the Pillar Spot (DI): Not very useful | 1 | 0
  A website/app to access APRETUDE information- the Pillar Spot (DI): Somewhat useful | 8 | 0
  A website/app to access APRETUDE information- the Pillar Spot (DI): Useful | 14 | 0
  A website/app to access APRETUDE information- the Pillar Spot (DI): Extremely useful | 7 | 0
  The website to access APRETUDE information (RI): number analyzed (Participants) | 0 | 25
  The website to access APRETUDE information (RI): Not at all useful | 0 | 1
  The website to access APRETUDE information (RI): Not very useful | 0 | 1
  The website to access APRETUDE information (RI): Somewhat useful | 0 | 6
  The website to access APRETUDE information (RI): Useful | 0 | 11
  The website to access APRETUDE information (RI): Extremely useful | 0 | 6

48. Secondary Outcome: Number of SSPs Assessed for Perceptions of Utility of Implementation Strategies and Facilitators and Barriers to Acceptability of RI and DI
Description: Perceptions of Utility of Implementation Strategies and Facilitators and Barriers to Acceptability of RI and DI measured from themes emerging from Proctor and CFIR guided semi-structured qualitative interview. In this outcome measure, SSPs provided their insights on the tools and strategies used for implementing APRETUDE during the PILLAR study.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on the SSPs who were interviewed and had data available for the specified analysis at the specified time points. All questions were not administered to both RI and DI arms; hence only participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 25 | 16
Participants
  Medication Administration Planner | 7 | 4
  Frequently Asked Questions (FAQs) | 11 | 8
  Readiness Considerations | 4 | 4
  Getting Started Overview | 4 | 11
  Injection Education Video | 13 | 10
  Drop-in visits (DI): number analyzed (Participants) | 25 | 0
  Drop-in visits (DI) | 11 | 0
  Designated injection days (DI): number analyzed (Participants) | 25 | 0
  Designated injection days (DI) | 5 | 0
  Prescheduled Appointments (DI): number analyzed (Participants) | 25 | 0
  Prescheduled Appointments (DI) | 18 | 0
  Transportation services (DI): number analyzed (Participants) | 25 | 0
  Transportation services (DI) | 10 | 0
  PrEP Communication Options Tool (DI): number analyzed (Participants) | 25 | 0
  PrEP Communication Options Tool (DI) | 8 | 0
  Implementation guidance video (DI): number analyzed (Participants) | 25 | 0
  Implementation guidance video (DI) | 10 | 0
  How to discuss sexual health guidance (DI): number analyzed (Participants) | 25 | 0
  How to discuss sexual health guidance (DI) | 3 | 0
  Acquisition Tracker (DI): number analyzed (Participants) | 25 | 0
  Acquisition Tracker (DI) | 1 | 0

49. Secondary Outcome: Number of PSPs Assessed for Perceptions of Utility of Implementation Strategies Through Semi-Structured Interviews (SSIs)
Description: Perceptions of Utility of Implementation Strategies and Facilitators and Barriers to Acceptability of RI and DI measured from themes emerging from Proctor and CFIR guided semi-structured qualitative interview. In this outcome measure, PSPs provided their insights regarding the tools and strategies used for delivering APRETUDE.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who completed an interview at the specified time point. All questions were not administered to both RI and DI arms; hence only participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 23 | 21
Participants
  Getting Started brochure | 10 | 9
  Participant handbook | 7 | 10
  Patient brochure | 7 | 12
  Patient website (RI): number analyzed (Participants) | 0 | 21
  Patient website (RI) | 0 | 11
  What to expect video (DI): number analyzed (Participants) | 23 | 0
  What to expect video (DI) | 13 | 0
  Myths facts video (DI): number analyzed (Participants) | 23 | 0
  Myths facts video (DI) | 9 | 0
  HIV education video (DI): number analyzed (Participants) | 23 | 0
  HIV education video (DI) | 11 | 0
  ViiV Connect Assistance Video (DI): number analyzed (Participants) | 23 | 0
  ViiV Connect Assistance Video (DI) | 6 | 0
  Reminder service text (DI): number analyzed (Participants) | 23 | 0
  Reminder service text (DI) | 7 | 0
  Appointment scheduler (DI): number analyzed (Participants) | 23 | 0
  Appointment scheduler (DI) | 5 | 0

50. Secondary Outcome: Number of Injections Occurring Within Target Window From Target Date
Description: This outcome measure evaluates the number of injections occurring within the target window. The target window is defined as ± 7 days from target date of injection for Dose 2 and subsequent injections.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Units; unit: Injections
Units Other Than Participants: Injections
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 111 | 81
Number analyzed (Injections) | 111 | 81
Injections
  Dose 2 | 103 | 76
  Dose 3: number analyzed (Participants) | 105 | 77
  Dose 3: number analyzed (Injections) | 105 | 77
  Dose 3 | 77 | 57
  Dose 4: number analyzed (Participants) | 99 | 72
  Dose 4: number analyzed (Injections) | 99 | 72
  Dose 4 | 66 | 49
  Dose 5: number analyzed (Participants) | 93 | 71
  Dose 5: number analyzed (Injections) | 93 | 71
  Dose 5 | 50 | 45
  Dose 6: number analyzed (Participants) | 88 | 67
  Dose 6: number analyzed (Injections) | 88 | 67
  Dose 6 | 44 | 30
  Dose 7: number analyzed (Participants) | 81 | 65
  Dose 7: number analyzed (Injections) | 81 | 65
  Dose 7 | 35 | 27
  Dose 8: number analyzed (Participants) | 1 | 1
  Dose 8: number analyzed (Injections) | 1 | 1
  Dose 8 | 0 | 0

51. Secondary Outcome: Number of PSPs Completing Target Number of Injections
Description: Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: as for outcome 50
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants | 81 | 63

52. Secondary Outcome: Number of PSPs With Perceptions of Facilitators to Fidelity to Injections
Description: Perceptions of utility of implementation strategies and facilitators and barriers to acceptability of RI and DI measured from themes emerging from Proctor and CFIR guided semi-structured qualitative interviews. In this outcome measure, PSPs provided their insights into how APRETUDE has been incorporated into their daily lives, including factors that supported its delivery.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 23 | 21
Participants
  APRETUDE Fitting life | 23 | 20
  Clinic staff supporting incorporation of APRETUDE into schedule | 15 | 10
  Booking appointments in advance | 13 | 11
  Easy to fit into life (convenience, etc.) | 16 | 8
  No transportation issues | 5 | 15
  Good fit with work schedule | 13 | 6
  Clinic hours aligned with patient schedule | 11 | 4

53. Secondary Outcome: Number of PSPs With Perceptions of Barriers to Fidelity to Injections
Description: Perceptions of utility of implementation strategies and facilitators and barriers to acceptability of RI and DI measured from themes emerging from Proctor and CFIR guided semi-structured qualitative interviews. In this outcome measure, PSPs reported several challenges related to incorporating APRETUDE into their daily lives.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 23 | 21
Participants
  Discomfort | 14 | 11
  Clinic challenges | 4 | 6
  Work challenges | 2 | 5

54. Secondary Outcome: Number of SSPs With Perceptions of Facilitators to Fidelity to Injections
Description: Perceptions of utility of implementation strategies and facilitators and barriers to acceptability of RI and DI measured from themes emerging from Proctor and CFIR guided semi-structured qualitative interviews. In this outcome measure, SSPs provided insights regarding the facilitators for adherence to APRETUDE and the support provided to enable patient adherence. These facilitators were categorized as resources, support, patient communication and patient feasibility.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 25 | 16
Participants
  Resources: Communication (call, email and text) | 7 | 2
  Resources: Dedicated injection nurse for follow-up | 2 | 3
  Resources: Patient education about importance of adherence | 1 | 4
  Resources: Dedicated support staff for each step: education, authorization, etc | 4 | 0
  Resources: Flexibility of using oral PrEP for bridging when needed | 1 | 3
  Support: Scheduling appointments in advance | 4 | 3
  Support: Team dedicated for follow-up | 5 | 1
  Patient Communication: Increasing global communication | 6 | 5
  Patient Communication: Encouraging proactively engaging patients with scheduling | 6 | 3
  Patient Communication: Accessibility for patients for open line communication | 8 | 2
  Patient feasibility: APRETUDE is feasible for patients | 9 | 3
  Patient feasibility: Clinical staff making the process run smoothly | 4 | 4
  Patient feasibility: Working around patient schedule helps with feasibility | 3 | 3

55. Secondary Outcome: Number of SSPs With Perceptions of Barriers to Fidelity to Injections
Description: Perceptions of utility of implementation strategies and facilitators and barriers to acceptability of RI and DI measured from themes emerging from Proctor and CFIR guided semi-structured qualitative interviews. In this outcome measure, SSPs provided insights regarding the barriers and challenges in enabling patient adherence to APRETUDE. The barriers were categorized as patient barriers and staff challenges.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 25 | 16
Participants
  Patient Barriers: Scheduling Barriers | 4 | 2
  Patient Barriers: Vulnerable Population | 2 | 2
  Patient Barriers: Traveling | 2 | 2
  Patient Barriers: Patients hard to contact (e.g., no phone access) | 2 | 2
  Staff Challenges: Concern about patients missing injection window | 4 | 2
  Staff Challenges: Not being able to contact patients who miss an appointment | 1 | 3

56. Secondary Outcome: Number of SSPs Who Administer Sexual Health Assessment (SHA)
Description: In this outcome measure, SSPs answered questions about their administration of the sexual health assessment (SHA). The SHA was only administered by SSPs at the DI sites, hence it was not assessed for RI sites.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP
Number analyzed (Participants) | 52
Participants
  Yes | 14
  No And Not Planning to Use the Sexual Health Assessment | 14
  No But Planning to Use the Sexual Health Assessment | 4
  I don't know | 20

57. Secondary Outcome: Number of Eligible PSPs for Which SHA Are Administered
Description: In this outcome measure, data shown below describes the number of PSPs to which the SHA was administered.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who completed at least one SHA survey at any timepoint. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  Yes | 39 | 35
  No | 15 | 13
  I don't know | 23 | 15
  Missing | 40 | 21

58. Secondary Outcome: Number of Men Who Have Sex With Men (MSM) and Transgender Men (TGM) Who Take the SHA Through M12
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach.
  Timeframe for evaluation of this outcome measure is M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: The protocol-defined endpoint for this outcome specifically requires data presentation by MSM and TGM, so data here are displayed by those groups. Data for this endpoint was collected from all MSM and TGM across DI and RI arms in alignment with the objective, therefore the analysis by MSM and TGM was not completed within arms but across arms.
Measure: Count of Participants; unit: Participants
Groups:
- Men Who Have Sex With Men (MSM): MSM who were HIV negative prior to initiation of CAB PrEP and who had either not received PrEP or were current or prior users of oral PrEP were included.
- Transgender Men (TGM): TGM who were HIV negative prior to initiation of CAB PrEP and who had either not received PrEP or were current or prior users of oral PrEP were included.
Arm/Group | Men Who Have Sex With Men (MSM) | Transgender Men (TGM)
Number analyzed (Participants) | 189 | 12
Participants
  Yes | 73 | 1
  No | 25 | 3
  I don't know | 36 | 2
  Missing | 55 | 6

59. Secondary Outcome: Number of MSM and TGM Who Report Having Had Sex in the Last 6 Months on the SHA
Description: In this outcome measure, data shown below describes the number of MSM and TGM who reported having had sex in the last 6 months.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: As pre-specified in the protocol, this outcome measure was evaluated in the MSM and TGM separately. Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who completed at least one SHA survey at any timepoint. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Men Who Have Sex With Men (MSM) | Transgender Men (TGM)
Number analyzed (Participants) | 189 | 12
Participants
  No | 5 | 1
  Yes | 128 | 5
  I prefer not to answer | 1 | 0
  Missing | 55 | 6

60. Secondary Outcome: Number of PSPs Who Expressed Interest in PrEP or Never Heard of PrEP Out of Those Who Report Having Had Sex in the Last 6 Months
Description: In this outcome measure, data presented below shows the number of PSPs who expressed interest in PreP by responding to the question "Have you taken oral PreP in the last 6 months" and number of PSPs who had not heard of PreP.
Time Frame: Up to Month 12
Population: as for outcome 57
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  Before enrolling in this study, you ever heard of people without HIV taking oral PrEP pills?: Yes | 70 | 61
  Before enrolling in this study, you ever heard of people without HIV taking oral PrEP pills?: No | 30 | 15
  Before enrolling in this study, you ever heard of people without HIV taking oral PrEP pills?: I don't know/prefer not to answer | 7 | 3
  Before enrolling in this study, you ever heard of people without HIV taking oral PrEP pills?: Missing | 10 | 5
  Before enrolling in this study, had you heard of APRETUDE?: Yes | 68 | 58
  Before enrolling in this study, had you heard of APRETUDE?: No | 39 | 21
  Before enrolling in this study, had you heard of APRETUDE?: I don't know/prefer not to answer | 0 | 0
  Before enrolling in this study, had you heard of APRETUDE?: Missing | 10 | 5
  Have you taken oral PrEP in the last 6 months?: Yes | 77 | 65
  Have you taken oral PrEP in the last 6 months?: No | 26 | 11
  Have you taken oral PrEP in the last 6 months?: I don't know/prefer not to answer | 2 | 1
  Have you taken oral PrEP in the last 6 months?: Missing | 12 | 7

61. Secondary Outcome: Number of PSPs Who Initiate APRETUDE After Taking the SHA
Description: In this outcome measure, PSPs were asked if they had taken oral PreP in the last 6 months. PSPs who answered 'No' or 'I prefer not to answer' were further asked if they had ever taken oral PreP.
  Timeframe for evaluation of this outcome measure is through M12(equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: as for outcome 57
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  Have you taken oral PrEP in the last 6 months?: Yes | 77 | 65
  Have you taken oral PrEP in the last 6 months?: No | 26 | 11
  Have you taken oral PrEP in the last 6 months?: I prefer not to answer | 2 | 1
  Have you taken oral PrEP in the last 6 months?: Missing | 12 | 7
  Have you ever taken oral PrEP: number analyzed (Participants) | 28 | 12
  Have you ever taken oral PrEP: Yes | 5 | 1
  Have you ever taken oral PrEP: No | 11 | 0
  Have you ever taken oral PrEP: I prefer not to answer | 1 | 0
  Have you ever taken oral PrEP: Missing | 11 | 11

62. Secondary Outcome: Number of PSPs With Perceptions of SHA
Description: Perceptions of the sexual health assessment (SHA) among PSPs were measured from themes emerging from Proctor and CFIR guided semi-structured qualitative interviews.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who completed an interview at the specified time point. This question was not administered to the RI arm; hence they were not assessed. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 23 | 0
Participants
  SHA was received by PSPs | 16 | 0
  SHA was not received by PSPs | 3 | 0
  SHA received/not received- Missing | 4 | 0
  SHA found useful by PSPs: number analyzed (Participants) | 16 | 0
  SHA found useful by PSPs | 15 | 0
  SHA not found useful by PSPs: number analyzed (Participants) | 16 | 0
  SHA not found useful by PSPs | 0 | 0
  SHA found useful/not useful- Missing: number analyzed (Participants) | 16 | 0
  SHA found useful/not useful- Missing | 1 | 0

63. Secondary Outcome: Number of SSPs With Perceptions of SHA
Description: In this outcome measure, SSPs provided insights regarding the use and implementation of SHA tool in their clinic/practice. The SHA was only administered by SSPs at the DI sites, hence it was not assessed for RI sites.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP
Number analyzed (Participants) | 18
Participants
  The Sexual Health Assessment is/will be easy to implement in my clinic/practice: Completely disagree | 1
  The Sexual Health Assessment is/will be easy to implement in my clinic/practice: Disagree | 1
  The Sexual Health Assessment is/will be easy to implement in my clinic/practice: Neither agree nor disagree | 3
  The Sexual Health Assessment is/will be easy to implement in my clinic/practice: Agree | 8
  The Sexual Health Assessment is/will be easy to implement in my clinic/practice: Completely agree | 5
  The Sexual Health Assessment is/will be an easy way to identify individuals interested in PrEP: Completely disagree | 1
  The Sexual Health Assessment is/will be an easy way to identify individuals interested in PrEP: Disagree | 0
  The Sexual Health Assessment is/will be an easy way to identify individuals interested in PrEP: Neither agree nor disagree | 3
  The Sexual Health Assessment is/will be an easy way to identify individuals interested in PrEP: Agree | 10
  The Sexual Health Assessment is/will be an easy way to identify individuals interested in PrEP: Completely agree | 4
  The Sexual Health Assessment helps/will help to facilitate conversations about PrEP with patients: Completely disagree | 1
  The Sexual Health Assessment helps/will help to facilitate conversations about PrEP with patients: Disagree | 0
  The Sexual Health Assessment helps/will help to facilitate conversations about PrEP with patients: Neither agree nor disagree | 3
  The Sexual Health Assessment helps/will help to facilitate conversations about PrEP with patients: Agree | 8
  The Sexual Health Assessment helps/will help to facilitate conversations about PrEP with patients: Completely agree | 6

64. Secondary Outcome: Number of Modifications Reported by SSPs Using FRAME-IS
Description: The Framework for Reporting Adaptations and Modifications to Evidence-based Implementation Strategies (FRAME-IS) is a measure that provides a precise understanding of modifications, the process of modifying or adapting, and the relationship between different forms of modification and subsequent health and implementation outcomes. Data below summarize all modifications reported by SSPs during PILLAR study.
  Timeframe for evaluation of this outcome measure is from M2 to M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: At Month 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: Analysis was performed on data submitted from SSPs who completed at least one FRAME-IS assessment at any time point and had data available for the specified analysis at the specified time points.
Measure: Number; unit: Number of Modifications
Arm/Group | DI- SSP | RI- SSP
Number analyzed (Participants) | 56 | 30
Number of Modifications
  Trial Month 2 Modifications | 6 | 3
  Trial Month 3 Modifications | 4 | 8
  Trial Month 4 Modifications | 3 | 0
  Trial Month 5 Modifications | 3 | 5
  Trial Month 6 Modifications | 4 | 3
  Trial Month 7 Modifications | 1 | 4
  Trial Month 8 Modifications | 3 | 2
  Trial Month 9 Modifications | 2 | 0
  Trial Month 10 Modifications | 10 | 0
  Trial Month 11 Modifications | 2 | 0
  Trial Month 12 Modifications | 5 | 1

65. Secondary Outcome: Number of Modifications for Each Category Reported by SSPs Using FRAME-IS
Description: The FRAME-IS is a measure that provides a precise understanding of modifications, the process of modifying or adapting, and the relationship between different forms of modification and subsequent health and implementation outcomes. Data below summarize the types of modifications and adaptations reported by SSPs during PILLAR study.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: as for outcome 64
Measure: Number; unit: Number of Modifications
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 56 | 30
Number of Modifications
  Content: Modification made to the content of APRETUDE materials and tools | 12 | 4
  Evaluation: Modification made to the staff evaluate whether APPRETUDE is working | 5 | 3
  Training: Modification made to the staff delivering APRETUDE are trained | 22 | 0
  Contextual: Modification made to the overall implementation of APRETUDE injection delivered | 30 | 22

66. Secondary Outcome: Number of Modifications Made for Adaptations to Implementation Reported by SSPs Using FRAME-IS
Description: The FRAME-IS is a measure that provides a precise understanding of modifications, the process of modifying or adapting, and the relationship between different forms of modification and subsequent health and implementation outcomes. Data below summarize the perceptions and motivations of adaptations to implementation reported by SSPs using FRAME-IS.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: as for outcome 64
Measure: Number; unit: Number of Modifications
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 56 | 30
Number of Modifications
  Increase the number of patients with access to APRETUDE | 23 | 5
  Improve feasibility of the implementation effort | 19 | 8
  Improve fit with the clinical/practice setting | 18 | 10
  Increase satisfaction with the implementation effort | 17 | 11
  Speed up injection/implementation process | 17 | 12

67. Secondary Outcome: Number of PSPs Assessed for Perceptions of Adaptations to Implementation Strategies
Description: PSP perceptions of adaptations to implementation strategies were measured from themes emerging from Proctor and CFIR guided semi-structured qualitative interviews. In this outcome measure, PSPs discussed their use of study resources and recommendations to staff for delivery of APRETUDE.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 23 | 21
Participants
  Discussed tools and resources | 21 | 20
  Positive feedback about tools and resources | 10 | 7
  Only used tools/resources in the beginning of PILLAR | 5 | 7
  Does not remember tools or resources | 3 | 5
  Resources were helpful | 2 | 4
  Negative feedback about tools and resources | 2 | 4
  Did not use (pay much attention to resources) | 2 | 2
  Recommendations to staff | 16 | 14
  Would not change anything | 4 | 3
  APRETUDE education within the community | 1 | 3
  Being culturally aware and non-judgmental | 2 | 2
  Support APRETUDE schedule | 2 | 1
  Discussion about post-Injection discomfort | 1 | 2

68. Secondary Outcome: Number of PSPs With History of PrEP Use That Complete the SHA and ISQ and Start APRETUDE
Description: In this outcome measure, PSPs who completed the SHA and ISQ, describe the history of PrEP use and of sexual health assessment use for determination of PreP use during PILLAR study.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who completed at least one ISQ and SHA survey at any timepoint. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 39 | 35
Participants
  Have you ever taken oral PrEP- Yes: number analyzed (Participants) | 28 | 12
  Have you ever taken oral PrEP- Yes | 5 | 1
  Have you ever taken oral PrEP- No: number analyzed (Participants) | 28 | 12
  Have you ever taken oral PrEP- No | 11 | 0
  Have you ever taken oral PrEP- Prefer not to answer: number analyzed (Participants) | 28 | 12
  Have you ever taken oral PrEP- Prefer not to answer | 1 | 0
  Have you ever taken oral PrEP- Missing: number analyzed (Participants) | 28 | 12
  Have you ever taken oral PrEP- Missing | 11 | 11
  The SHA asked questions to determine if PrEP was right for me- Completely disagree | 2 | 1
  The SHA asked questions to determine if PrEP was right for me- Disagree | 0 | 1
  The SHA asked questions to determine if PrEP was right for me- Neither agree nor disagree | 5 | 7
  The SHA asked questions to determine if PrEP was right for me- Agree | 19 | 11
  The SHA asked questions to determine if PrEP was right for me- Completely Agree | 13 | 15

69. Secondary Outcome: Number of PSPs With Reasons for Choosing and Switching to APRETUDE Assessed by Semi-Structured Interviews (SSIs)
Description: Reasons for choosing and switching to APRETUDE were measured from themes emerging from Proctor and CFIR guided semi-structured qualitative interviews among PSPs. In this outcome measure, PSPs shared previous oral PrEP experiences, comparisons of other forms of PrEP to APRETUDE, and reasons for preferring APRETUDE.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on all PSPs who were administered at least one dose of APRETUDE injection or of CAB tablets for PrEP and who completed an interview at the specified time point. Only those participants with data available for the specified analysis at the specified time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 23 | 21
Participants
  Oral PrEP used: Challenges remembering to take pill every day | 16 | 11
  Oral PrEP used: Side effects of oral PrEP | 6 | 3
  APRETUDE differences to oral PrEP: Better adherence and feeling more protected | 4 | 5
  APRETUDE differences to oral PrEP: APRETUDE More convenient than Oral | 6 | 2
  APRETUDE differences to oral PrEP: Less/ No side effects related to oral PrEP | 0 | 5
  Prefer APRETUDE over Oral PrEP: More convenient | 14 | 8
  Prefer APRETUDE over Oral PrEP: Less/No side effects | 1 | 5

70. Secondary Outcome: Number of PSPs With Reasons for Choosing and Switching to APRETUDE Assessed by ISQs
Description: The ISQ uses a variety of questions to assess outcomes spanning acceptability of, feasibility of, utility of, and experiences with the intervention and the implementation approach. In this outcome measure, PSPs answered ISQ regarding reasons for choosing to take APRETUDE.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 117 | 84
Participants
  I want a prevention option that is more convenient for my life | 66 | 49
  I won't have to remember to take PrEP everyday | 63 | 45
  I do not have to worry or stress about missing a dose like oral PrEP | 55 | 47
  I want to try a new approach and see if it fits into my life | 43 | 27
  I will not have to worry about HIV every day | 43 | 27

71. Secondary Outcome: Number of PSPs Assessed for Perception of Facilitators
Description: General perceptions of facilitators for APRETUDE delivery and use were measured among PSPs from themes emerging from Proctor and CFIR guided semi-structured qualitative interviews. In this outcome measure, PSPs discuss views of long-term use of APRETUDE, reasons to choose APRETUDE, and experiences with clinic staff.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 23 | 21
Participants
  Would consider APRETUDE as a long-term treatment | 19 | 17
  APRETUDE as long-term treatment provides protection | 12 | 6
  APRETUDE as long-term treatment provides peace of mind | 4 | 6
  APRETUDE as long-term treatment has concerns about insurance coverage long-term | 4 | 3
  APRETUDE as long-term treatment has convenience over oral PrEP | 5 | 1
  APRETUDE as long-term treatment taken as long as necessary | 0 | 5
  Reasons others may choose APRETUDE: Convenience and ease of use | 8 | 3
  Reasons others may choose APRETUDE: Health and prevention | 4 | 5
  Global judgement of recommend to others | 13 | 14
  Experiences of care: Discussed interactions with clinic staff | 21 | 21
  Experiences of care: Clinic staff were friendly and kind | 17 | 19
  Experiences of care: PSP was treated with respect | 15 | 15
  Experiences of care: Clinic staff were knowledgeable | 12 | 7
  Experiences of care: Shared decision making | 10 | 9
  HIV/STI testing: Testing frequency was acceptable | 13 | 15
  HIV/STI testing: Positive experience with scheduling HIV/ STI testing | 11 | 11
  Reported whether they discussed APRETUDE with family / friends | 21 | 18
  Has discussed APRETUDE with partner(s) | 11 | 9
  Peers have started PrEP | 10 | 7
  Uptake of PrEP by Friends | 3 | 2

72. Secondary Outcome: Number of PSPs Assessed for Perception of Barriers
Description: General perceptions of barriers for APRETUDE delivery and use were measured among PSPs from themes emerging from Proctor and CFIR guided semi-structured qualitative interviews. In this outcome measure, PSPs discuss challenging views of or experiences with APRETUDE receipt.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for PSPs who received OLI).
Time Frame: Up to Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
Number analyzed (Participants) | 23 | 21
Participants
  Would not consider APRETUDE as a long-term treatment | 1 | 3
  Cost Challenges | 6 | 3
  Challenges with switching insurance carriers | 0 | 4

73. Secondary Outcome: Number of SSPs Assessed for Perception of Facilitators
Description: General perceptions of facilitators for APRETUDE intervention and implementation were measured among SSPs from themes emerging from Proctor and CFIR guided semi-structured qualitative interviews. In this outcome measure, SSPs discuss clinic culture and implementation motivations.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on the SSPs who were interviewed and had data available at the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 25 | 16
Participants
  Supportive leadership for implementation | 11 | 11
  Leadership willing to help/support | 6 | 8
  Leadership being actively involved in the process | 4 | 5
  APRETUDE positively accepted | 10 | 5
  Team adaptability | 8 | 3
  Staff being supportive of the clinic offering APRETUDE | 11 | 6
  Aiming to improve patient's health | 2 | 2

74. Secondary Outcome: Number of SSPs Assessed for Perception of Barriers
Description: General perceptions of barriers for APRETUDE intervention and implementation were measured among SSPs from themes emerging from Proctor and CFIR guided semi-structured qualitative interviews. In this outcome measure, SSPs discuss feelings and perspectives while implementing APRETUDE.
  Timeframe for evaluation of this outcome measure is through M12 (equivalent to M13 for SSPs who assessed PSPs receiving OLI).
Time Frame: Up to Month 12
Population: Analysis was performed on the SSPs who were interviewed and had data available at the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | DI - SSP | RI - SSP
Number analyzed (Participants) | 25 | 16
Participants
  Staff having mixed feelings | 9 | 4
  Initial negative response due to extra workload | 2 | 2

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were reported from signing of informed consent (a period starting up to 90 days before the first dose in Month 1) to Month 12 (study completion). Non serious Drug related AEs were reported from Month 1 (first dose) to Month 12 (study completion).
Description: Month 12 (study completion) is equivalent to Month 13 for PSPs who received OLI and for SSPs who assessed PSPs receiving OLI. Adverse events for SSPs were not collected as it was not required as per study design.
Arm/Group | Dynamic Implementation (DI) - PSP | Routine Implementation (RI) - PSP
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/84
Serious Adverse Events (participants affected / at risk) | 1/117 | 0/84
Other Adverse Events (participants affected / at risk) | 5/117 | 6/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dynamic Implementation (DI) - PSP (N=117) | Routine Implementation (RI) - PSP (N=84)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dynamic Implementation (DI) - PSP (N=117) | Routine Implementation (RI) - PSP (N=84)
Injection site pain (General disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 2 (2) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT05374525/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT05374525/SAP_001.pdf